### ALDER BIOPHARMACEUTICALS, INC.

#### **Clinical Trial Protocol**

Clinical Trial Title A Parallel Group, Double-Blind, Randomized, Placebo

Controlled Phase 3 Trial to Evaluate the Efficacy and Safety of ALD403 Administered Intravenously in

Patients with Chronic Migraine

Protocol Number ALD403-CLIN-011

Investigational Product ALD403

Indication Treatment for the Prevention of Chronic Migraine

Sponsor Alder BioPharmaceuticals, Inc.

11804 North Creek Pkwy S Bothell, WA 98011 USA Phone: +1 425-205-2900 Fax: +1 425-205-2901

Sponsor's Medical Monitor

Alder BioPharmaceuticals, Inc.

Phone:

Clinical Trial Compliance This clinical trial will be conducted in accordance with

standards of Good Clinical Practice, as defined by the International Conference on Harmonisation and all

applicable federal and local regulations.

EudraCT No. 2016-001306-41

Date of Protocol (original release) 17-Aug-2016
Date of Amendment 1 24-Oct-2016
Date of Amendment 2 20-Mar-2017
Date of Amendment 3 31-Aug-2017

#### **Confidential Information**

The confidential information in this document is provided to you as an Investigator, potential Investigator, or Consultant, for review by you, your staff, and applicable institutional review committees. This information will not be disclosed to others without written authorization from Alder BioPharmaceuticals, Inc., except to the extent necessary to obtain informed consent from those persons to whom the drug may be administered.

#### SIGNATURE PAGE

## **Declaration of Sponsor**

Title: A Parallel Group, Double-Blind, Randomized, Placebo Controlled Phase 3 Trial to Evaluate the Efficacy and Safety of ALD403 Administered Intravenously in Patients with Chronic Migraine

This clinical trial protocol was subject to critical review. The information it contains is consistent with current knowledge of the risks and benefits of the Investigational Product, with moral ethical and scientific principles governing clinical research, and in accordance with Good Clinical Practice and applicable federal and local regulations.



VP, Clinical Development Alder BioPharmaceuticals, Inc.



Principal Investigator

#### DECLARATION OF THE PRINCIPAL INVESTIGATOR

Title: A Parallel Group, Double-Blind, Randomized, Placebo Controlled Phase 3 Trial to Evaluate the Efficacy and Safety of ALD403 Administered Intravenously in Patients with Chronic Migraine

This clinical trial protocol was subject to critical review. The information it contains is consistent with current knowledge of the risks and benefits of the Investigational Product, with moral ethical and scientific principles governing clinical research, and in accordance with Good Clinical Practice and applicable federal and local regulations.

| Timelparinvesugator | |
|---------------------|-------------|
| Signature | |
| Name (printed) | |
| Title | |
| Institution | <del></del> |

# 1. PROTOCOL SYNOPSIS

| Title | A Parallel Group, Double-Blind, Randomized, Placebo<br>Controlled Phase 3 Trial to Evaluate the Efficacy and Safety of<br>ALD403 Administered Intravenously in Patients with Chronic<br>Migraine |
|---|---|
| Sponsor | Alder BioPharmaceuticals, Inc. |
| Investigational Product | ALD403, a humanized anti-(calcitonin gene-related peptide) (CGRP) monoclonal antibody |
| Primary Objective | To evaluate the efficacy of repeat doses of ALD403 administered intravenously (IV) compared to placebo in patients with chronic migraine. |
| Secondary Objectives | To evaluate the safety of repeat doses of ALD403 administered IV compared to placebo in patients with chronic migraine. To evaluate the pharmacokinetics (PK) and immunogenicity of repeat doses of ALD403 administered IV to patients with chronic migraine. |
| Methodology | This will be a parallel group, double-blind, randomized, placebo-<br>controlled trial. Subjects will be randomized into one of two<br>ALD403 dose levels (100 mg or 300 mg) or placebo in a 1:1:1<br>ratio. Randomization will be stratified by baseline migraine days<br>(<17 and ≥17 days during screening) and prophylactic medication<br>use during 3 months prior to screening (prophylactic medication<br>use vs. no prophylactic medication use). |
| | Visits will occur at screening, randomization (on-site or phone), Day 0, and Weeks 2, 4, 8, 12, 16, 20, 24, and 32. Subjects will complete the eDiary daily through Week 24. Eligible subjects will be randomized 28 to 30 days after the screening visit, and treated (first dose) on Day 0, 0-8 days after the randomization visit. Treatment includes two infusions of ALD403 or placebo administered on Days 0 and 84 (Week 12). Subjects will be followed for 20 weeks after the final dose for total study duration of approximately 36 weeks, including the screening period. |
| Number of Subjects<br>Planned | Approximately 1050 subjects will be randomized and treated at approximately 150 centers in the US and worldwide. |
| Subject Selection Criteria | Males and females between 18 and 65 years of age, inclusive, who were diagnosed with migraines at $\leq 50$ years of age, and have a history of chronic migraine for $\geq 12$ months before screening. During the 28 day screening period, subjects must complete the headache eDiary 24 out of 28 days and must have |

| | 11.1 |
|---|---|
| | headaches occurring on $\geq 15$ to $\leq 26$ days of which at least 8 must be migraine days. |
| Investigational Product, | There will be 3 treatment groups of approximately 350 subjects |
| Dose and Schedule | each. Subjects will receive IV infusions of the assigned treatment on Day 0 and on Day 84. |
| | 1. 100 mg ALD403<br>2. 300 mg ALD403 |
| | 3. Placebo |
| Duration of Treatment | Two doses of ALD403/placebo will be given 12 weeks apart |
| Duration of Clinical Trial | The trial participation period will be approximately 36 weeks. |
| Participation | This will include a 4 week screening period, a 12 week treatment |
| | period and a 20 week follow-up period. |
| Clinical Trial Endpoints | Primary Efficacy Endpoint: |
| | • Change in frequency of migraine days (Weeks 1-12) |
| | Key Secondary Endpoints: |
| | • 75% migraine responder rate (Weeks 1-4) |
| | • 75% migraine responder rate (Weeks 1-12) |
| | • 50% migraine responder rate (Weeks 1-12) |
| | Percentage of subjects with a migraine on the day after |
| | dosing |
| | • Reduction in migraine prevalence from baseline to Week 4 |
| | Other Secondary Endpoints: |
| | Headaches/migraines with acute medication usage |
| | Acute migraine medication usage |
| | • Change in frequency of migraine days (Weeks 1-24) |
| | • 100% migraine responder rate (Weeks 1-12) |
| | <ul> <li>Migraine responder rates for time periods other than Weeks<br/>1-12</li> </ul> |
| | • Change in frequency of migraine days between baseline and |
| | time periods other than Weeks 1-12 |
| | Headache responder rates Change in the frequency of headache days. |
| | <ul><li>Change in the frequency of headache days</li><li>Percent change in headache or migraine days</li></ul> |
| | <ul> <li>Time to first migraine after dosing</li> </ul> |
| | Headache/migraine hours |
| | Headache/migraines with severe intensity |
| | <ul> <li>Patient Global Impression of Change (PGIC)</li> </ul> |
| | • Short-Form Health Survey (SF-36) |
| | <ul> <li>Health-Related Quality of Life (EQ-5D-5L)</li> </ul> |
| | Headache Impact Test (HIT-6) |

#### **Tertiary Endpoints**

- Headache episodes/migraine attacks
- Migraine symptom-free days
- Most Bothersome Symptom (MBS)

#### Safety Endpoints

- Adverse events (AEs) and serious adverse events (SAEs)
- Clinical laboratory assessments
- Vital signs
- Electrocardiograms (ECGs)
- Columbia-Suicide Severity Rating Scale (C-SSRS)

#### Pharmacokinetic and Immunogenicity Endpoints

- Free ALD403 plasma concentrations
- Development of specific anti-ALD403 antibodies
- Characterization of specific anti-ALD403 antibodies for neutralizing activity

#### **Concomitant Medications**

Concomitant medications must be recorded in the Case Report Form (CRF).

Barbiturates and prescription opiates are allowed for  $\leq 4$  days per month through Week 24, provided the subject has been on a stable regimen ( $\leq 4$  days per month) for at least 2 months prior to screening.

Any botulinum toxin injections for migraine or for any other medical/cosmetic reasons are prohibited within 4 months prior to screening and during the study through Week 24.

Devices, neuromodulation, neurostimulation, or injectable therapy (trigger point injections) for headache prophylaxis are prohibited 2 months prior to screening and during the study through Week 24.

Monoamine oxidase inhibitors (MAOIs), ketamine, methysergide, methylergonovine, and nimesulide are prohibited within 3 months prior to screening and during the study through Week 24.

Other medications taken for headache prophylaxis will be permitted provided that the dose has been stable for at least 3 months prior to screening and there are no alterations to their regimen through Week 24.

#### Sample Size

1050 subjects will be randomized into 3 treatment groups in a balanced ratio (approximately 350/group). Pair-wise testing of

| | each ALD403 group vs. placebo will be performed using a 5% two-sided alpha level. Three hundred and fifty subjects per group provides at least 90% power for the primary endpoint assuming a treatment effect of at least 1 day and a common standard deviation of 4 days or less. For the key secondary 75% responder rate endpoints 90% power is achieved for the pair-wise comparisons, assuming a placebo responder rate of 20%, and an ALD403 rate of 31%. |
|---|---|
| Statistical Analysis | Efficacy and safety endpoints will be summarized with descriptive statistics. |
| | Statistical inferential testing of the primary efficacy endpoint and key secondary endpoints will be performed while maintaining a |
| | study wide type-I error rate of two sided 5%. The primary |
| | analyses will test for a difference between the active treatment groups and placebo in Weeks 1-12, change in frequency of |
| | migraine days. The primary analyses will be based on ANCOVA |
| | model. The migraine responder rates and percentage of subjects with a migraine on the day after dosing will be tested with |
| | stratified Cochran Mantel Haenszel (CMH) tests. The same |
| | stratification factors as used in randomization will be used to |
| | perform these tests. Repeated measures will be used to test for the reduction in migraine prevalence from baseline to Week 4. |
| | The migraine days reported during the initial 28-days of |
| | screening will be used as baseline. Following treatment, migraine data will be summarized and analyzed in 28 day |
| | intervals (e.g. Weeks 1-4, 5-8, 9-12). The change from baseline |
| | in migraine days for a given 4-week interval will be the difference between migraine days in that interval and the |
| | migraine days during baseline. The Week 1-12 change from |
| | baseline measure, for a subject, will be the average of the change |
| | from baseline results from each of the three intervals. A 75% responder, for a given 4-week interval, will be a subject |
| | with a $\geq 75\%$ reduction in migraine days during that interval. A |
| | 75% responder over Weeks 1-12 will be a subject who achieves average reduction of $\geq$ 75% over this time period based upon the |
| | Week 1-12 change from baseline measure. Subjects who do not |
| Dharmacolzinatia Analysia | complete their eDiary will have their missing data imputed. |
| Pharmacokinetic Analysis | The concentrations of ALD403 will be measured in plasma from all ALD403 treated subjects using a validated assay method. |
| | The PK analysis of plasma will include determination of the free ALD403 concentrations at the following times: Day 0 (within 1 hour before dosing), immediately post-dose (within 15 minutes of end of infusion), Weeks 2, 4, 8, 12 (within 1 hour before dosing), 24, and 32. |

For subjects receiving placebo, selected samples will be analysed.

Blood specimens will be collected for the detection of anti-ALD403 antibody, and when appropriate the samples will be analysed also for neutralizing anti-ALD403 antibody activity on Day 0 (pre-dose within 1 hour before dosing), Weeks 2, 4, 8, 12 (within 1 hour before dosing), 24, and 32. Subjects who test positive for specific anti-ALD403 antibodies at the time of the last study visit will be asked to provide additional blood samples for immunogenicity testing.

#### 2. SCHEDULE OF EVENTS AND ASSESSMENTS

| Assessment | Screen | Rand <sup>1</sup> 28-30 days after Screen | Day 0 <sup>2</sup> Tx within 8 days after Rand | Week 2<br>Day 14<br>-3 days | Week 4<br>Day 28<br>± 3 days | Week 8<br>Day 56<br>± 3 days | Week 12<br>Day 84<br>±3 days<br>Tx | Week 16<br>Day 112<br>± 3 days | Week 20<br>Day 140<br>± 3 days | Week 24<br>Day 168<br>+7 days <sup>3</sup> | Week 32<br>EOS/ET<br>Day 224<br>± 7 days |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Informed Consent | X | | | | | | | | | | |
| Inclusion/Exclusion Criteria Review | X | X | X | | | | | | | | |
| Demographics | X | | | | | | | | | | |
| Medical History | X | | | | | | | | | | |
| Headache eDiary Data Review and Compliance Check <sup>4</sup> | X | X | X | X | X | X | X | X | X | X | |
| Headache eDiary closeout <sup>5</sup> | | | | | | | | | | X | X |
| Height and Weight <sup>6</sup> | X | | X | | | | X | | | X | X |
| Physical Exam <sup>7</sup> | X | | X | | | | X | | | X | X |
| Patient Global Impression of Change (PGIC) | | | | | X | X | X | X | X | X | X |
| Most Bothersome Symptom (MBS) | X | | X | | X | X | X | X | X | X | X |
| Vital Signs <sup>8</sup> | X | | X | | X | X | X | X | X | X | X |
| C-SSRS <sup>9,10</sup> | X | | X | X | X | X | X | X | X | X | X |
| 12-lead ECG <sup>11</sup> | X | | X | | | | X | | | | X |
| Hematology, Chemistry <sup>12</sup> | X | | X | | | | X | | | | X |
| Serology (HIV, Hepatitis B and C) | X | | | | | | | | | | |
| Urine Drugs Abuse Screen | X | | | | | | | | | | |
| Urine Pregnancy (hCG) Test <sup>10</sup> | X | | X | | | | X | | | | X |
| Plasma ALD403 (PK) <sup>12</sup> | | | X | X | X | X | X | | | X | X |
| Serum Anti-ALD403 Ab <sup>12</sup> | | | X | X | X | X | X | | | X | X |
| SF-36, EQ-5D-5L, and HIT-6 | X | | X | | X | | X | X | | X | X |
| AE Review | X | X | X | X | X | X | X | X | X | X | X |
| Concomitant Medication Review | X | X | X | X | X | X | X | X | X | X | X |
| Randomization | | X | | | | | | | | | |
| ALD403/placebo administration <sup>13</sup> | | | X | 0.0 1 /5 1 | | | X | | | | |

Abbreviations: TX: Treatment, Rand: Randomization, EOS/ET: End of Study/Early Termination Please refer to next page for footnotes.

- <sup>1</sup> Randomization will occur 28-30 days after the screening visit after eligibility assessments are approved by the Medical Monitor and eligibility, including eDiary eligibility criteria, are confirmed by the investigator. Every effort should be made to conduct an on-site randomization visit; however, a phone visit is acceptable in cases where the subject's schedule will not permit an on-site visit.
- <sup>2</sup> Dosing must occur within 8 days after randomization.
- <sup>3</sup> Week 24 visit must be done on the target day or seven days after. The visit may not be conducted earlier than the target date.
- <sup>4</sup> Headache eDiary distributed at the screening visit. eDiary review and compliance check through Week 24.
- <sup>5</sup> eDiary closeout must be performed at Week 24, or at the ET visit while the subject is on site.
- <sup>6</sup> Height and weight collected at screening visit. Weight only collected on Day 0 (pre-dose) and at Weeks 12 (pre-dose), 24, and 32 or ET.
- <sup>7</sup> Physical exam must be done pre-dose on Day 0 and Week 12.
- <sup>8</sup> Vital signs measured pre-dose and within 2 hours post-dose on Days 0 and Week 12.
- <sup>9</sup> C-SSRS "Baseline/Screening Version" should be used at screening, and C-SSRS "Since Last Visit Version" should be used on Day 0 (pre-randomization), Weeks 2,4, 8, 12 (pre-dose), 16, 20, 24, and 32 or ET.
- <sup>10</sup>Inclusion/exclusion criteria review, C-SSRS, and urine pregnancy test must be done prior to dosing on Day 0. C-SSRS and urine pregnancy test must be done prior to dosing at Week 12.
- <sup>11</sup>Conduct ECG pre-dose, and within 2 hours post dose on Day 0 and Week 12.
- <sup>12</sup>Blood draws obtained pre-dose on dosing days (within 1 hour before dosing). On Day 0, draw additional PK immediately post dose (within 15 minutes of end of infusion). Subjects who test positive for anti-ALD403 antibodies at the last study visit will be asked to provide up to 2 additional blood samples for immunogenicity testing at 3 month intervals for up to 6 months.
- <sup>13</sup>Subjects must be monitored for at least 2 hours after the dosing completion to assess for the occurrence of adverse events. Subjects will be requested to stay longer than 2 hours after dosing should the investigator determine this is clinically warranted (e.g., subjects should be observed until all AEs are resolved or clinically stable).

#### 3. LIST OF ABBREVIATIONS

AE Adverse event

ADL Activities of Daily Living
ALP Alkaline phosphatase
ALT Alanine aminotransferase
ANCOVA Analysis of Covariance
AST Aspartate aminotransferase

AUC Area under the concentration-time curve

BMI Body Mass Index BP Blood pressure

CGRP Calcitonin Gene-Related Peptide

CRF Case Report Form

C-SSRS Columbia-Suicide Severity Rating Scale

DMC Data Monitoring Committee

DNA Deoxyribonucleic acid
EC Ethics Committee
ECG Electrocardiogram

EDC Electronic Data Capture

EQ-5D-5L Health-Related Quality of Life

ET Early Termination

FDA Food and Drug Administration

GCP Good Clinical Practice
HIT-6 Headache Impact Test
IB Investigator's Brochure

ICD International Classification of Diseases

ICF Informed Consent Form

ICH International Conference on Harmonization

ICHD International Classification of Headache Disorders

IHS International Headache Society

IgG1 Immunoglobulin G1
IP Investigational Product
IRB Institutional Review Board

IV Intravenous

IWRS Interactive Web Response System

Kg Kilogram

LLOQ Lower Limit of Quantification

M Molarity

m2 Meter squared

mAb Monoclonal antibody

MAOI Monoamine oxidase inhibitor
MBS Most Bothersome Symptom
MCH Mean corpuscular hemoglobin

MCHC Mean corpuscular hemoglobin concentration

MCV Mean corpuscular volume

MedDRA Medical Dictionary for Regulatory Activities

mg Milligram
mL Milliliter
mm Millimeter

MRM Menstrually-related migraine
NOAEL No-observed-adverse-effect-level
NSAID Non-steroidal anti-inflammatory drug

PK Pharmacokinetic

PGIC Patient Global Impression of Change QTcF QT corrected using Fridericia formula

RBC Red blood cell

SAE Serious adverse event
SF-36 Short Form Health Survey
TMD Temporomandibular Disorder

WBC White blood cell

# 4. TABLE OF CONTENTS

| ALDER | BIOPHARMACEUTICALS, INC. | 1 |
|--------|----------------------------------------------|----|
| SIGNAT | ΓURE PAGE | 2 |
| DECLA | RATION OF THE PRINCIPAL INVESTIGATOR | 3 |
| 1. | PROTOCOL SYNOPSIS | 4 |
| 2. | SCHEDULE OF EVENTS AND ASSESSMENTS | 9 |
| 3. | LIST OF ABBREVIATIONS | 11 |
| 4. | TABLE OF CONTENTS | 13 |
| 5. | INTRODUCTION | 17 |
| 5.1. | Investigational Product | 17 |
| 5.2. | Background | 17 |
| 5.3. | Investigational Product | 19 |
| 5.3.1. | Summary of Nonclinical Studies | 19 |
| 5.3.2. | Summary of Clinical Trials | 21 |
| 5.3.3. | Dose Justification. | 22 |
| 5.4. | Risks and Benefits | 22 |
| 5.5. | Compliance Statement | 23 |
| 6. | OBJECTIVES | 24 |
| 6.1. | Primary Objective | 24 |
| 6.2. | Secondary Objectives | 24 |
| 7. | TRIAL DESIGN | 25 |
| 7.1. | Clinical Trial Endpoints | 25 |
| 7.1.1. | Primary Efficacy Endpoint | 25 |
| 7.1.2. | Key Secondary Endpoints: | 25 |
| 7.1.3. | Other Secondary Endpoints: | 25 |
| 7.1.4. | Tertiary Endpoints | 26 |
| 7.1.5. | Safety Endpoints | 26 |
| 7.1.6. | Pharmacokinetic and Immunogenicity Endpoints | 26 |
| 7.2. | Clinical Trial Design. | 26 |
| 7.3. | Data Monitoring Committee | 27 |
| 7.4. | Methods to Minimize/Avoid Bias | 27 |
| 8 | SELECTION AND WITHDRAWAL OF SUBJECTS | 28 |

| 8.1. | Inclusion Criteria | 28 |
|---------|-----------------------------------------------------------|----|
| 8.2. | Exclusion Criteria | 29 |
| 8.3. | Registration and Treatment Assignment | 32 |
| 8.3.1. | Registration Procedure, Subject Numbering | 32 |
| 8.3.2. | Randomization and Treatment Assignment | 32 |
| 8.4. | Subject Treatment Discontinuation and Early Withdrawal | 33 |
| 8.4.1. | Criteria for Discontinuation from Study Treatment | 33 |
| 8.4.2. | Criteria for Withdrawal from the Clinical Trial | 33 |
| 8.4.3. | Timing of Withdrawal | 32 |
| 8.4.4. | Follow-up for Early Withdrawal | 32 |
| 8.4.5. | Replacement Policy | 32 |
| 8.4.6. | Lost to Follow-Up | 32 |
| 9. | CLINICAL TRIAL TREATMENTS | 35 |
| 9.1. | Investigational Product | 35 |
| 9.2. | Placebo | 35 |
| 9.3. | Investigational Product Dosing and Administration | 35 |
| 9.3.1. | Packaging and Labeling. | 36 |
| 9.3.2. | Blinding | 36 |
| 9.3.3. | Storage and Handling of Investigational Product | 36 |
| 9.3.4. | Accountability and Disposition of Investigational Product | 37 |
| 9.4. | Concomitant Medications | 37 |
| 10. | STUDY ASSESSMENTS AND PROCEDURES | 39 |
| 10.1. | Schedule of Assessments | 39 |
| 10.2. | Assessments and Procedures | 39 |
| 10.2.1. | Randomization | 39 |
| 10.2.2. | Demographics | 39 |
| 10.2.3. | Medical History | 39 |
| 10.2.4. | Physical Examinations | 40 |
| 10.2.5. | Vital Signs | 40 |
| 10.2.6. | Questionnaires | 41 |
| 10.2.7. | Columbia-Suicide Severity Rating Scale (C-SSRS) | 41 |
| 10.2.8. | Most Bothersome Symptom (MBS) | 41 |
| 10.2.9. | Other Questionnaires | 42 |

| 10.2.10. | 12-Lead ECG | 42 |
|---|---|---|
| 10.2.11. | Laboratory Samples and Testing | 42 |
| 10.3. | eDiary Completion and Compliance Review | 43 |
| 11. | ASSESSMENT OF SAFETY | 45 |
| 11.1. | Adverse Events | 45 |
| 11.1.1. | Definitions | 45 |
| 11.1.2. | Assessment of Adverse Events | 45 |
| 11.1.3. | Recording Adverse Events | 47 |
| 11.1.4. | Reporting Serious Adverse Events | 48 |
| 11.1.5. | Unexpected and Related Serious Adverse Events | 49 |
| 11.1.6. | Follow-up of Adverse Events | 50 |
| 11.1.7. | Clinical Laboratory Tests | 50 |
| 11.1.8. | Pregnancy | 50 |
| 11.1.9. | Suicidal Ideation and Behavior | 51 |
| 11.2. | Management of Reactions to ALD403 | 51 |
| 12. | ASSESSMENT OF EFFICACY, PHARMACOKINETICS, AND IMMUNOGENICITY | 53 |
| 12.1. | Efficacy | 53 |
| 12.1.1. | eDiary | 53 |
| 12.1.2. | Endpoints | 53 |
| 12.2. | Pharmacokinetics | 57 |
| 12.3. | Immunogenicity | 57 |
| 13. | STATISTICAL CONSIDERATIONS | 59 |
| 13.1. | Decision Rule | 59 |
| 13.2. | Sample Size | 59 |
| 13.3. | General Considerations | 59 |
| 13.3.1. | Definition of Baseline | 59 |
| 13.3.2. | Handling of Missing Data | 59 |
| 13.3.3. | Populations to be Analyzed | 60 |
| 13.4. | Statistical Methods | 60 |
| 13.4.1. | Subject Disposition, Demographics and Baseline Characteristics | 61 |
| 13.4.2. | Efficacy Analyses | 61 |
| 13.4.3. | Analysis of Drug Concentrations | 63 |

| 13.4.4. | Safety Analyses | 63 |
|---|---|---|
| 14. | ETHICAL, LEGAL AND ADMINISTRATIVE ASPECTS | 65 |
| 14.1. | Data Quality Assurance | 65 |
| 14.2. | Case Report Forms and Source Documents | 65 |
| 14.3. | Study Documentation | 65 |
| 14.4. | Data Collection and Electronic Data Capture (EDC) | 65 |
| 14.5. | Archiving Clinical Trial Records | 66 |
| 14.6. | Good Clinical Practice | 66 |
| 14.7. | Informed Consent | 67 |
| 14.8. | Protocol Approval and Amendment | 67 |
| 14.8.1. | Premature Termination of the Clinical Trial | 68 |
| 14.9. | Confidentiality | 68 |
| 14.10. | Publication Policy | 68 |
| 15. | APPENDICES | 70 |
| 15.1. | Migraine preventive therapies with established or probable efficacy <sup>17,18,19</sup> | 70 |
| 15.2. | Columbia-Suicide Severity Rating Scale (C-SSRS) Risk Assessment | 71 |
| 15.2.1. | Baseline/Screening Version | 71 |
| 15.2.2. | Since Last Visit Version | 74 |
| 15.3. | Headache Impact Test (HIT-6 v1.0) | 77 |
| 15.4. | Short-Form Health Survey (SF-36 v2.0) | 78 |
| 15.5. | Health Related Quality of Life (EQ-5D-5L) | 82 |
| 15.6. | Patient Global Impression of Change (PGIC) | 85 |
| 15.7. | Most Bothersome Symptom (MBS) | 86 |
| 15.8. | References | 87 |

#### 5. INTRODUCTION

# 5.1. Investigational Product

ALD403 is a humanized anti-(calcitonin gene-related peptide) (CGRP) monoclonal antibody (anti-CGRP) that is being developed by Alder BioPharmaceuticals, Inc., for the prophylaxis of migraine.

# 5.2. Background

Migraine is a highly prevalent paroxysmal neurological disease characterized by recurrent episodes of moderate to severe headache associated with physiological disruptions of neurological, gastrointestinal, and sensory function. Episodes typically last between 4 and 72 hours and recur often without warning over decades of time. It is most prevalent through the 3<sup>rd</sup> and 4<sup>th</sup> decades of life with a significant gender bias of 3:1 for women. Migraine is the most prevalent neurological disease for which medical treatment is sought, and considered the 6th leading cause of disability in the world. Annually, lost work time and diminished productivity attributable to migraine costs American employers an estimated \$19.6 billion.

Migraine appears to have a significant genetic/epigenetic component to its etiology and it is observed in all age groups, races, and ethnicities. Generally, migraine begins as an episodic disease. Between episodes of migraine the nervous system returns to a normal (premorbid) state of function. However, approximately 2.5% of people with episodic migraine will annually transform from episodic to chronic migraine, meaning they are experiencing migraine on greater than 15 days per month for at least 3 consecutive months. For those with chronic migraine, the headaches are more intense; migraine-associated symptoms, more severe; and the disease-related impact and disability are much greater than observed for episodic migraine. In addition, chronic migraine is associated with more co-morbid diseases such as anxiety, depression, and non-headache pain.

The pathophysiology of migraine is complex and incompletely understood. Current models of migraine are based on a genetically determined hyper-excitable nervous system characterized by a lowered threshold to sensory activation and uniqueness in its sensory processing.<sup>7</sup> Interactions between this migraine nervous system and specific internal and external stimuli (migraine triggers) can result in activation of the trigeminovascular system (TVS). Once activated the TVS

releases various vasoactive peptides generating peripheral sensitization of trigeminal and upper cervical nociceptors. The ensuing peripheral nociceptive stimuli synapse in the Trigeminal Nucleus Caudalis to ultimately create a state of central sensitization. Clinically, this process is observed as a fully developed attack of migraine.

Central to this model of migraine is calcitonin gene-related peptide (CGRP). CGRP is one of the most abundant peptides in the human body and is produced in both peripheral and central neurons. It is abundant in trigeminal neurons and when released is involved in the vasodilation, inflammatory cascade, and pain transmission associated with migraine. In both peripheral and central pain pathways CGRP is associated with pain transmission and neuronal sensitization. Intravenous (IV) infusions of CGRP can cause a migraine-like headache in susceptible individuals with migraine. In addition, many pharmacological agents used as acute or prophylactic treatment of migraine are known to inhibit CGRP. Thus CGRP is an attractive target for development of novel migraine pharmacology.

Currently the pharmacological treatment of migraine can be divided into acute treatment, that is, medications designed to reverse a migraine after it is initiated and preventive treatment that is designed to protect the nervous system from generating migraine. Acute treatments are used intermittently only as needed to stop an attack while preventative treatments are used on a sustained basis for periods of month to years. Acute treatment while generally quite effective can actually worsen the severity and frequency of migraine when used too frequently, a condition called medication overuse headache (MOH).<sup>4</sup> MOH is common in populations with frequent episodic and chronic migraine.<sup>11</sup>

Numerous medications are used to prevent migraine but to date none have been designed specifically for migraine. These commonly include tricyclic antidepressants, beta-blockers, and certain anticonvulsants. It is estimated that 45% of adults with frequent episodic migraine and virtually all with chronic migraine would benefit from effective preventive medications yet only an estimated 12% of this population are currently using a migraine preventive. In large measure, this is due to poor tolerability, lack of efficacy, and failure to adhere to treatment. Clearly there is a medical need to develop effective, well-tolerated and safe preventive treatments for migraine.

# 5.3. Investigational Product

ALD403 is a genetically engineered humanized immunoglobulin G1 (IgG1) antibody that binds to human-α-CGRP with an affinity of 1.5E-11 M and human-β-CGRP with an affinity of 5.7E-11 M.

## 5.3.1. Summary of Nonclinical Studies

A nonclinical testing program has been conducted supporting the use of ALD403 in clinical trials. More detailed discussion is provided in the current version of the ALD403 Investigator's Brochure (IB).

ALD403 is a genetically engineered humanized IgG1 antibody that binds to  $\alpha$ - and  $\beta$ - forms of human, cynomolgus monkey, and rat CGRP. The amino acid sequence for  $\alpha$ - and  $\beta$ -CGRP is identical in cynomolgus monkeys and humans (data on file); therefore the *in vitro* binding characteristics of cynomolgus monkey and human CGRP to ALD403 would be indistinguishable. Rat  $\alpha$ -CGRP is one amino acid different from human  $\alpha$ -CGRP and rat  $\beta$ -CGRP is 3 amino acids different from human  $\beta$ -CGRP. Based on comparable binding affinity and *in vitro* potency for rat, cynomolgus monkey, and human  $\alpha$ - and  $\beta$ -CGRP, the rat and cynomolgus monkey were selected for nonclinical safety assessments.

Pharmacodynamic activity by ALD403 in the species selected for toxicological investigations (rats, rabbits, and monkeys) was confirmed in vivo by conducting studies to determine the ability of ALD403 to inhibit CGRP-mediated neurogenic dermal vasodilation.

In the single-dose nonclinical toxicology studies, the no-observed-adverse-effect-level (NOAEL) for IV administration of ALD403 to rats and cynomolgus monkeys was 100 mg/kg.

Toxicological investigations in rats and monkeys indicated that repeated-dose IV of ALD403 at 10, 30, or 100 mg/kg once weekly for four weeks was well tolerated, with no signs of adverse effects related to treatment. Under the conditions of these studies, the no-observed-adverse-effect-level (NOAEL) for once weekly IV administration of ALD403 to rats or monkeys for four weeks was 100 mg/kg.

A chronic multiple-dose toxicology study in cynomolgus monkeys was conducted to evaluate the potential effects by ALD403 following 6-months administration via slow bolus injection once

every two weeks (a total of fourteen dosing occasions) at 0, 20, 50, or 150 mg/kg/dose followed by a three month recovery period in select animals.

Following the sixth dosing occasion on study day 71, one low-dose (20 mg/kg/dose) female animal exhibited an anaphylactoid-like reaction and died within approximately 30 minutes. Collectively, the clinical, gross, and microscopic findings were consistent with an ADA-mediated anaphylactoid event as the cause of death. Humanized monoclonal antibodies are known for their potential to illicit severe immunologic reactions in monkeys and therefore, the death of one animal was considered as a class effect.

Administration of ALD403 via intravenous (slow bolus) injection once every 2 weeks for approximately 6-months (for a total of 14 doses) did not result in any treatment-related effects upon the parameters evaluated in this study. The NOAEL for ALD403 following chronic administration in monkeys was considered to be 150 mg/kg/dose (Day 183 mean  $C_{max}$  of 19,600/6,160  $\mu$ g/mL; mean AUC  $_{(0\text{-}2wk)}$  of 1,610,000/904,000  $\mu$ g·h/mL for males/females, respectively).

ALD403 is not expected to interact directly with DNA or other chromosomal materials, and genotoxicity assessments have not been conducted. The carcinogenic potential for ALD403 has not been thoroughly investigated. The results of toxicological and clinical investigations to date with ALD403 have provided no indications of effects with the potential to support or induce the proliferation of malignant cells.

Definitive embryo-fetal development studies with ALD403 in rats and rabbits have been conducted. The administration of ALD403 by intravenous (slow bolus) injection to pregnant female rats on Days 6, 12 and 18 post coitum or pregnant female New Zealand White rabbits on Days 7, 13 and 20 post coitum, at 75 or 150 mg/kg/dose was well tolerated, and there was no evidence of embryo-fetal mortality (embryolethality), alterations in growth (fetotoxicity), or structural abnormalities (teratogenicity) in either species.

The local tolerance of ALD403 was assessed following repeated-(once weekly) dose studies in rats and cynomolgus monkeys utilizing ALD403 administered IV. Following the end-of-treatment, no gross or microscopic lesions were observed in the ALD403 injection sites excised from rats. In the injection sites obtained from cynomolgus monkeys, only procedure-related findings were observed and included (in order of decreasing incidence) minimal and/or mild

superficial perivascular infiltrates, fibroplasia/fibrosis, myointimal hyperplasia of the injected vein, hemorrhage, and sporadic observations in the epidermis and skeletal muscle.

# **5.3.2.** Summary of Clinical Trials

Detailed descriptions of the relevant clinical findings for ALD403 are provided in the Investigator's Brochure (IB).

A summary of completed and ongoing ALD403 clinical trials is shown in Table 5.3

**Table 5.3 ALD403 Clinical Trials** 

| Trial ID | Phase/Objective | Trial Subject<br>Population | Total<br>Number of<br>Subjects in<br>the Trial | Number of<br>Subjects<br>Randomized<br>and Dosed with<br>ALD403 | Number of<br>Subjects<br>Randomized<br>and Dosed<br>with Placebo |
|---|---|---|---|---|---|
| ALD403-CLIN-001 (completed) | Phase 1<br>Safety | Healthy<br>Volunteer <sup>1</sup> | 104 | 67 | 37 |
| ALD403-CLIN-002<br>(completed) | Phase 1b<br>Safety & Efficacy | Frequent<br>Episodic<br>Migraine | 163 | 81 | 82 |
| ALD403-CLIN-003<br>(completed) | Phase 1<br>Safety | Healthy<br>Volunteer | 60 | 36 | 24 |
| ALD403-CLIN-005 <sup>2</sup> (completed) | Phase 2<br>Safety & Efficacy | Chronic Migraine | 616 | 495 | 121 |
| ALD403-CLIN-006 <sup>2</sup> (ongoing) | Phase 3 Safety & Efficacy | Frequent<br>Episodic<br>Migraine | 888 | 666 | 222 |
| ALD403-CLIN-007<br>(completed) | Phase 1<br>Safety | Healthy<br>Volunteer | 60 | 49 | 11 |
| ALD403-CLIN-009<br>(completed) | Phase 1<br>Safety | Healthy<br>Volunteer | 36 | 24 | 12 |
| ALD403-CLIN-010 (completed) | Phase 1<br>Safety | Healthy<br>Volunteer | 24 | 16 | 8 |
| ALD403-CLIN-012 <sup>3</sup> (ongoing) | Phase 1<br>Safety | Type 1 Diabetic (T1DM) | 21 | 14 | 7 |
| ALD403-CLIN-013 <sup>3</sup> (ongoing) | Phase 3<br>Safety, Open<br>Label | Chronic Migraine | 128 | 128 | |

<sup>&</sup>lt;sup>1</sup> ALD403-CLIN-001 included a subset of seven migraine subjects.

<sup>&</sup>lt;sup>2</sup> Enrollment in this blinded clinical trial has been completed and subjects are in the follow-up phase of the trial.

<sup>&</sup>lt;sup>3</sup> Enrollment in this open label clinical trial has been completed and subjects are in the follow-up phase of the trial.

#### **5.3.3.** Dose Justification

ALD403 doses of 100 and 300 mg met the primary efficacy endpoint through Week 12 post-treatment across a number of measures and had an acceptable safety profile in a prior phase 2 trial, ALD403-CLIN-005. Therefore, these doses were selected for this study to be administered every 12 weeks.

#### 5.4. Risks and Benefits

ALD403 may prevent migraine from occurring in patients treated in this trial. No specific toxicities or adverse effects related to the blockade of CGRP by ALD403 have been identified in either the nonclinical toxicology program or the clinical trials with ALD403 that have been completed to date.

There may be unknown adverse effects and unforeseeable risks associated with study drug administration or unexpected interactions with another drug that have not yet been identified.

As with all protein therapeutics, there is a risk of a serious allergic reaction. In completed ALD403 trials conducted to date, no serious allergic reactions have been observed with the administration of ALD403 in humans.

In the completed ALD403 clinical trials with headache patients, the most common observed adverse events (>5%) with receiving ALD403 or placebo included upper respiratory tract infection, back pain, dizziness, arthralgia, urinary tract infection, and headache. The majority of these adverse events were categorized as mild to moderate.

Long term data with ALD403 is limited.

- Healthy volunteer trials have included limited dosing, short duration of follow up and have not include long term follow-up.
- Trials in migraine patients have also included limiting dosing. These trials are currently
  ongoing and no new significant findings have been noted during the follow-up period to
  date.

The safety findings to date indicate that ALD403 Injection is well tolerated, and demonstrates a favorable benefit-risk profile based on review of nonclinical, clinical, and scientific literature data.

# **5.5.** Compliance Statement

This clinical trial will be conducted in accordance with standards of Good Clinical Practice (GCP) as defined by the International Conference on Harmonisation (ICH) and all applicable federal and local regulations.

# 6. **OBJECTIVES**

# 6.1. Primary Objective

The primary objective is:

To evaluate the efficacy of repeat doses of ALD403 administered IV compared to placebo in patients with chronic migraine.

# 6.2. Secondary Objectives

The secondary objectives include the following:

- To evaluate the safety of repeat doses of ALD403 administered IV compared to placebo in patients with chronic migraine.
- To evaluate the pharmacokinetics (PK) and immunogenicity of repeat doses of ALD403 administered IV to patients with chronic migraine.

#### 7. TRIAL DESIGN

# 7.1. Clinical Trial Endpoints

Detail regarding the clinical trial endpoints and their derivation can be found in Section 12.1. Migraine headaches are defined as migraines as outlined in the International Headache Society (IHS) International Classification of Headache Disorders (ICHD, 3<sup>rd</sup> edition, beta version 2013), Section 1.3.<sup>4</sup> The presence or absence of aura will not impact the classification of a headache as a migraine.

# 7.1.1. Primary Efficacy Endpoint

• Change in frequency of migraine days (Weeks 1-12)

# 7.1.2. Key Secondary Endpoints:

- 75% migraine responder rate (Weeks 1-4)
- 75% migraine responder rate (Weeks 1-12)
- 50% migraine responder rate (Weeks 1-12)
- Percentage of subjects with a migraine on the day after dosing
- Reduction in migraine prevalence from baseline to Week 4

### 7.1.3. Other Secondary Endpoints:

- Headaches/migraines with acute medication usage
- Acute migraine medication usage
- Change in frequency of migraine days (Weeks 1-24)
- 100% migraine responder rate (Weeks 1-12)
- Migraine responder rates for time periods other than Weeks 1-12
- Change in frequency of migraine days between baseline and time periods other than Weeks 1-12
- Headache responder rates
- Change in the frequency of headache days
- Percent change in headache or migraine days
- Time to first migraine after dosing
- Headache/migraine hours

- Headache/migraines with severe intensity
- Patient Global Impression of Change (PGIC)
- Short-Form Health Survey (SF-36)
- Health-Related Quality of Life (EQ-5D-5L)
- Headache Impact Test (HIT-6)

#### 7.1.4. Tertiary Endpoints

- Headache episodes/migraine attacks
- Migraine symptom-free days
- Most Bothersome Symptom (MBS)

#### 7.1.5. Safety Endpoints

- Adverse events (AEs) and serious adverse events (SAEs)
- Clinical laboratory assessments
- Vital signs
- Electrocardiograms (ECGs)
- Columbia-Suicide Severity Rating Scale (C-SSRS)

#### 7.1.6. Pharmacokinetic and Immunogenicity Endpoints

- Free ALD403 plasma concentrations
- Development of specific anti-ALD403 antibodies
- Characterization of specific anti-ALD403 antibodies for neutralizing activity

# 7.2. Clinical Trial Design

This is a parallel group, double-blind, randomized, placebo-controlled trial of two infusions of ALD403 or placebo in patients with chronic migraine. Subjects who provide informed consent will be evaluated for eligibility based upon the inclusion and exclusion criteria.

Eligible subjects will be randomized 28-30 days after the screening visit and treated (first dose) on Day 0, within 8 days after the randomization visit. Treatment includes two infusions of ALD403 or placebo administered on Days 0 and 84 (Week 12). Subjects will be followed for 20 weeks after the final dose for total study duration of approximately 36 weeks, including the screening period.

Approximately 1050 subjects will be randomized and treated. Efficacy, safety, pharmacokinetic, and immunogenicity assessments will be conducted according to the Schedule of Events presented in Section 2.

# 7.3. Data Monitoring Committee

A Data Monitoring Committee (DMC) of qualified members will be formed to review trial data generated during the clinical trial. These members will not be otherwise affiliated with the Sponsor, and will not be connected with management of the clinical trial.

The primary focus of the DMC will be the safety of the clinical trial subjects. Based on the reviews and assessments of the data, the DMC will inform the Sponsor of any safety concerns and provide recommendations about stopping, modifying, or continuing the clinical trial. The DMC may also advise the Sponsor on the validity of continuing the trial and the scientific merit of the clinical trial. The DMC is not tasked with stopping the study early for efficacy or futility. DMC reviews will be conducted periodically throughout the study as outlined in the DMC Charter.

#### 7.4. Methods to Minimize/Avoid Bias

To minimize bias, this clinical trial is randomized, double-blinded, and placebo controlled. At the point of infusion, there are no obvious differences between ALD403 and placebo, and there are no known ALD403-specific safety or tolerability signals that could potentially unblind subjects and clinical trial staff. ALD403 is expected to have a fairly substantial impact on migraine frequency; however, the placebo effect in migraine studies is also reasonably large. Therefore, reduction in migraines is insufficient to deduce treatment assignment.

#### 8. SELECTION AND WITHDRAWAL OF SUBJECTS

#### 8.1. Inclusion Criteria

A subject must meet all of the following criteria during the screening period and on Day 0 to be eligible for inclusion in the trial:

- 1. Willing and able to read, understand, and sign the Informed Consent Form (ICF) and Assent Form for the clinical trial approved by the Investigator's local Review Board or a central Institutional Review Board (IRB) or Ethics Committee (EC).
- 2. Has adequate venous access for administration of investigational product and collection of blood samples.
- 3. Male or female 18-65 years of age, inclusive, at time of informed consent.
- Diagnosis of migraine at ≤ 50 years of age with history of chronic migraine ≥ 1 year prior to screening.
- 5. Prescription or over-the-counter medication for acute and/or prophylactic treatment of migraine has been prescribed or recommended by a healthcare professional.
- During the 28 day screening period, must have ≥ 15 to ≤ 26 headache days, of which ≥ 8 days were assessed as migraine days as documented in the eDiary (ICHD-III beta version, 2013 Section 1.3<sup>4</sup>).
- 7. Women of child-bearing potential, and males with partners of child-bearing potential, must agree to use adequate contraception for the duration of the study (from screening through Week 32) and for 6 months after the last dose of study drug. The following types of contraception are considered adequate provided they are locally authorized for use: oral, transdermal, or injectable (depot) estrogen and/or progestogen, selective estrogen receptor modulator therapy, intrauterine contraceptive device, double barrier method (e.g., condom and diaphragm or spermicidal gel) or vasectomy. Non-childbearing potential is defined as post-menopausal for at least 1 year, or surgical sterilization or hysterectomy at least 3 months before screening.
- 8. Any hormonal therapy (e.g., contraceptives, hormone replacement therapy) use is stable and ongoing for at least 3 months prior to screening.

- 9. Willing, committed, and able to comply with scheduled clinic visits and complete all trial-related procedures.
- 10. Headache eDiary was completed on at least 24 of the 28 days prior to randomization.
- 11. Any prophylactic use of medications for headaches must be stable for at least 3 months prior to screening.
- 12. Limited use of barbiturates (including Fiorinal®, Fioricet®, or any other combination containing butalbital) or prescription opiates (including single ingredient or combinations containing opiates, opioids, tramadol or tapentadol) by maintaining a stable dose for 2 months prior to screening and dosing is not expected to exceed 4 days per month through Week 24.
- 13. Subject agrees not to post any personal medical data or information related to the trial on any website or social media site (e.g., Facebook, Twitter) during the trial.
- 14. Subject is willing to complete the daily eDiary for the duration of the study and agrees to use the eDiary devices for the sole purpose of the ALD403-CLIN-011 study without alteration.

## 8.2. Exclusion Criteria

A subject who meets any of the following criteria will be excluded from the trial:

- 1. Confounding and clinically significant pain syndromes (e.g. fibromyalgia, chronic low back pain, complex regional pain syndrome).
- 2. Psychiatric conditions that are uncontrolled and/or untreated, including conditions that are not controlled for a minimum of 6 months prior to screening. Patients with a lifetime history of psychosis, mania, or dementia are excluded.
- 3. Diagnosis of acute or active temporomandibular disorders (TMD).
- 4. History or diagnosis of chronic tension-type headache, hypnic headache, cluster headache, hemicrania continua, new daily persistent headache, or unusual migraine subtypes such as hemiplegic migraine (sporadic and familial), ophthalmoplegic migraine and migraine with neurological accompaniments that are not typical of migraine aura (e.g., diplopia, altered consciousness, or long duration).

- 5. Any use of approved devices, neuromodulation, neurostimulation or injectable therapy (trigger point injections, extracranial nerve blocks, facet joint injections) are prohibited 2 months prior to screening and during the screening period.
- 6. Any use of botulinum toxin for migraine or for any other medical/cosmetic reasons requiring injections within 4 months prior to screening and during the screening period.
- 7. Any use of monoamine oxidase inhibitors (MAOIs), ketamine, methysergide, methylergonovine, or nimesulide within 3 months prior to screening or during the screening period.
- 8. Have present or previous malignancies, except:
  - Squamous or basal skin cell carcinoma with excision without evidence of recurrence
  - Malignancy  $\geq 10$  years since diagnosis/treatment without evidence of recurrence
- 9. Subject with known history or evidence of arteriosclerosis, cardiomyopathy, coronary artery disease, serious heart rhythm abnormalities, cerebrovascular disease, diabetes, Raynaud's disease, hereditary fructose intolerance, life-threatening allergy (e.g., anaphylaxis), or any active, progressive, or unstable cardiovascular, neurological, or autoimmune disorder. If questions arise, the Investigator should contact the Medical Monitor for guidance.
- 10. Clinically significant abnormal ECG during the screening period or on Day 0.
- 11. Any clinically significant concurrent medical condition or clinically significant laboratory abnormality during the screening period or on Day 0.
- 12. Body Mass Index (BMI)  $\geq$  39 kg/m<sup>2</sup> at screening.
- 13. Primary hypertension that is uncontrolled or newly diagnosed (systolic BP of > 139 mm Hg or diastolic BP of >89 mm Hg) at screening or secondary hypertension. Mild primary hypertension that is well-controlled for ≥ 6 months prior to screening is allowed.
- 14. The subject is at risk of self-harm or harm to others in the Investigator's opinion, based on clinical interview and responses provided on the Columbia-Suicide Severity Rating

- Scale (C-SSRS). Subjects must be excluded if they have a lifetime history of a serious suicide attempt or multiple suicide attempts (i.e., actual, interrupted, or aborted attempts), have had any suicidal behavior in the past 5 years (i.e., preparatory acts or behavior), or have had suicidal ideation of Type 3, 4, or 5 (i.e., suicidal ideation with any method without intent to act or suicidal ideation with intent to act, with or without a plan) in the past 6 months, as measured by the C-SSRS at Screening or on Day 0.
- 15. Any history or evidence of substance abuse or dependence (e.g., alcohol, opiates, amphetamines and barbiturates) within the past 2 years according to the International Classification of Diseases (ICD) 10: F10-19<sup>12</sup>
- 16. Pregnant, breastfeeding, or planning to become pregnant during the trial.
- 17. Receipt of any experimental, unregistered therapy (within or outside a clinical trial) within 30 days or 5 plasma half-lives (whichever is longer) before screening.
- 18. Receipt of any monoclonal antibody treatment (within or outside a clinical trial) within 6 months before screening.
- 19. Previously dosed with ALD403 or any monoclonal antibody targeting the CGRP pathway.
- 20. Planned or current participation in any other clinical trial during the duration of this clinical trial, or within 6 months before screening.
- 21. Recent or planned surgery, requiring general anesthesia, within 8 weeks prior to screening and during the duration of this clinical trial.
- 22. Positive for HIV, hepatitis B surface antigen, or hepatitis C antibody at screening.
- 23. Any condition that, in the opinion of the Investigator, would make the subject unsuitable for the clinical trial.
- 24. Employees of the Sponsor, CRO, or any clinical trial site involved in this trial and their immediate family members (i.e., parents, spouse, siblings, children).

# 8.3. Registration and Treatment Assignment

#### 8.3.1. Registration Procedure, Subject Numbering

Each participating investigative site will be assigned a 3-digit site number (e.g., 101, 102). At the screening visit, once the subject signs the ICF they are registered in the Interactive Web Response System (IWRS), which will assign a unique subject number. The first three digits of the subject number identify the site, and the remaining digits identify the subject.

Subjects who fail screening may be rescreened if approved in advance by the Medical Monitor.

## 8.3.2. Randomization and Treatment Assignment

Randomization will occur 28-30 days after the screening visit after eligibility assessments are approved by the Medical Monitor and eligibility, including eDiary criteria, are reconfirmed by the investigator.

Every effort should be made to conduct an on-site randomization visit, however a phone visit is acceptable in cases where the subject's schedule will not permit an on-site visit. Sites will complete randomization in IWRS, and the randomization assignment will be obtained by the clinical trial site's unblinded pharmacist or designee. Subjects will be randomized in equal ratios to one of the treatment groups. Stratified permuted block randomization will be used. Stratification will be by migraine days during the screening period (<17 days vs. ≥17 days) and prophylactic medication use during the 3 months prior to screening (prophylactic medication use vs. no prophylactic medication use).

Prophylactic medication use for migraine will be determined at screening based upon the subjects' medical history. Stratification for prophylactic medication use will be defined as any migraine preventive therapies listed in Appendix 15.1 that have been taken as a stable regimen for 3 months prior to screening. Use of other medications taken for migraine prophylaxis that are not listed in Appendix 15.1 will not be considered when determining stratification by prophylactic medication use.

Randomized subjects who terminate their clinical trial participation for any reason, regardless of whether Investigational Product was taken or not, will retain their randomization assignment and subject number.

# 8.4. Subject Treatment Discontinuation and Early Withdrawal

Subjects may discontinue treatment or withdraw from the clinical trial at any time and for any reason without penalty or prejudice to his or her future medical care.

## 8.4.1. Criteria for Discontinuation from Study Treatment

Study treatment must be discontinued for the following reasons:

- Pregnancy
- Suicidal ideation with intent, with or without a plan (i.e., 'yes' to suicidal ideation questions 4 or 5) or any suicidal behavior as determined by the C-SSRS.

Subjects discontinued due to suicidal ideation and or suicidal behavior must be referred to a mental health specialist as specified in Section 11.1.9.

Study treatment may also be discontinued for the following reasons:

- Adverse Event
- Subject decision
- Investigator decision
- Termination of the study by the Sponsor

If a subject discontinues study treatment due to a medical condition, Investigators must provide adequate medical treatment during study visits. Prior to removing a subject from study treatment, the decision should be discussed with the Sponsor Medical Monitor or designee. The reason for discontinuation from study treatment must be recorded on the CRF. Subjects who discontinue study treatment will be encouraged to continue with study assessments until the end of the study.

#### 8.4.2. Criteria for Withdrawal from the Clinical Trial

Subjects will be withdrawn from the clinical trial for any of the following reasons:

- Withdrawal of consent for the collection of clinical trial data including further access to medical records. The reason for withdrawal of consent will be recorded.
- Termination of the trial by the Sponsor
- Investigator decision
- Lost to follow-up

The reason for withdrawal and the date of withdrawal must be recorded on the CRF.

# 8.4.3. Timing of Withdrawal

Subjects are considered withdrawn from the clinical trial at the time that any of the criteria listed in Section 8.4.2 are met and the last study assessment is performed.

# 8.4.4. Follow-up for Early Withdrawal

Subjects who wish to withdraw their consent from study participation will be asked to have an early termination visit with associated visit assessments (see Schedule of Events in Section 2). Subjects who withdraw consent after randomization but do not receive study treatment may discontinue the study without any further procedures.

#### 8.4.5. Replacement Policy

Subjects who are withdrawn from the clinical trial after randomization will not be replaced, including subjects who withdraw between randomization and treatment. However, the target sample size is based upon the number of subjects randomized and treated.

#### 8.4.6. Lost to Follow-Up

If the subject fails to attend scheduled study visits or to respond to requests for follow-up, the clinical trial site will send a registered letter, at a minimum, to the subject requesting contact with the clinic. All attempts to resume contact (including copies of written correspondence and documentation of telephone and email contact attempts) will be included in the source documentation. Subjects who do not respond to requests for follow-up after all reasonable attempts to establish contact will be considered lost to follow-up.

#### 9. CLINICAL TRIAL TREATMENTS

# 9.1. Investigational Product

ALD403 is an anti-(calcitonin gene-related peptide) humanized monoclonal antibody (anti-CGRP mAb) that is being developed by Alder BioPharmaceuticals, Inc., for the prevention of migraine.

ALD403 Injection, 100 mg/vial, is presented in 2-mL Type I glass vials as a single-use preservative-free solution for IV administration. ALD403 is formulated at a concentration of 100 mg/mL with a pH of 5.8. Those subjects randomized to the ALD403 treatment group will receive an IV infusion of ALD403 Injection in 100 mL of 0.9% saline.

#### 9.2. Placebo

Placebo will be supplied as a single-use preservative-free solution in a 2-mL Type I glass vial formulated with the same excipients as ALD403, without the active ingredient. Those subjects randomized to placebo will receive an IV infusion Placebo in 100 mL of 0.9% saline.

# 9.3. Investigational Product Dosing and Administration

The pharmacist or designee responsible for receiving, storing, preparing and dispensing ALD403 and placebo IV infusions will be unblinded and will not be responsible for other aspects of the clinical trial where blinding is necessary. Dosing must occur within 8 days after randomization. Doses of ALD403 or placebo (total volume of 100 mL) will be administered IV over a period of 30 (+15) minutes on Day 0 and Week 12 (Day  $84 \pm 3$  days) by the blinded Investigator or designee (infusions may be administered for a total duration of up to 1 hour, if needed, in the judgement of the Investigator).

If the subject experiences a headache or migraine on dosing day and has no other clinically significant findings on Day 0, dosing may occur if it does not compromise the safety of the subject in the judgment of the Investigator. The Medical Monitor may be consulted as needed. Subjects must remain in the care facility and be monitored by site staff for at least 2 hours post-dose. The Investigator or sub-investigator must be immediately available during the infusion and for at least 2 hours post-dose to assess each subject for the occurrence of adverse events. Subjects will be requested to stay longer than 2 hours after dosing should the investigator determine this is clinically warranted (e.g., subjects should be observed until all AEs are resolved

or clinically stable). The timeframe for the post-dose observation period must be documented in the source record.

Further instructions on preparation and procedures associated with administering the IV can be found in the Pharmacy Manual.

## 9.3.1. Packaging and Labeling

Before the shipment to the investigative sites, Investigational Product (IP) will be labeled with information required by regulatory agencies, such as a statement that it is limited to investigational use. Investigational Product to be administered to the subject will be labeled by the site after dose preparation by the unblinded pharmacist or designee in a manner that protects blinding.

### 9.3.2. Blinding

This clinical trial is double-blinded, meaning the subjects and site personnel are blinded to treatment assignment, except for the clinical trial site's unblinded pharmacist or designee. The study site must have a written plan in place to ensure blinding is adequately maintained for the study. If the blind is broken, the date, time, and reason must be recorded. The blind should only be broken for reasons in which knowledge of the treatment assignment is critical to the management of subject safety. The Principal Investigator will report any cases of unblinding to the Sponsor within 24 hours of the incident.

#### 9.3.3. Storage and Handling of Investigational Product

Investigational Product/Placebo will be stored at a central depot or at the clinical site at -20°C (-10°C to -25°C) in accordance with any accompanying instructions. Please refer to the Pharmacy Manual for additional storage and handling procedures. Diluent (0.9% saline) will be stored according to manufacturer instructions.

Investigators shall take adequate precautions, including storage of the Investigational Product and Placebo in a securely locked, substantially constructed cabinet or other securely locked, substantially constructed enclosure, access to which is limited to maintain blind, prevent theft or diversion of the substance into illegal channels of distribution.
# 9.3.4. Accountability and Disposition of Investigational Product

The Investigator is responsible for maintaining accurate Investigational Product accountability records throughout the clinical trial. The site must maintain an Investigational Product Accountability Log as instructed in the Pharmacy Manual. Where more than one secure area is being used for storage at a site, all movement of Investigational Product through the chain of custody must be recorded in accountability records such that full reconciliation may be completed at the end of the trial.

Included with each Investigational Product shipment is a form listing lot numbers and quantity shipped. The Investigator, responsible pharmacist, or designee, will sign and return to Alder BioPharmaceuticals, Inc., or designee, a statement that certifies the receipt and integrity of these supplies. A copy will be retained for the site clinical trial file.

After completion of the clinical trial, the Investigator is responsible for either returning or destroying all unused Investigational Product. The Investigator must verify that no remaining supplies are in his/her possession. All used/partially used vials/IV bags will be destroyed onsite according to the site SOPs, or returned according to Alder BioPharmaceuticals, Inc. directive. Destruction must be in accordance with local regulations for the product type.

If the clinical trial is terminated, suspended, discontinued, or completed, the Investigator or designee shall return the unused supplies to the Sponsor or designee, or otherwise provide for disposition of the unused supplies (as authorized by the Sponsor).

### 9.4. Concomitant Medications

Any concomitant therapy used from the time the subject signs the informed consent form through Week 32 must be recorded on the eCRF, including medications required for treatment of any AEs or SAEs. The medication name, dosage, date, and indication for use must be recorded. The Medical Monitor or designee should be notified in advance of (or as soon as possible after) any instances in which restricted therapies are administered.

The following medications are **restricted** through Week 24:

Barbiturates and prescription opiates are allowed for ≤ 4 days per month through Week
 24, provided the subject has been on a stable regimen (≤ 4 days per month) for at least 2 months prior to screening.

- Any botulinum toxin injections for migraine or for any other medical/cosmetic reasons are prohibited within 4 months prior to screening and during the trial through Week 24.
- Devices, neuromodulation, neurostimulation, or injectable therapy (trigger point injections) for headache prophylaxis are prohibited 2 months prior to screening and during the trial through Week 24.
- Monoamine oxidase inhibitors (MAOIs), ketamine, methysergide, methylergonovine, and nimesulide are prohibited within 3 months prior to screening and during the trial through Week 24.

Any hormonal therapy (e.g., contraceptives, hormone replacement therapy) use must be stable for 3 months prior to screening and remain stable during the trial through Week 32.

Medications taken for headache prophylaxis will be permitted provided that the dose has been stable for at least 3 months prior to screening and there are no alterations to their regimen through Week 24. In general, changes to prophylactic headache medications during the trial are not allowed through Week 24. At the discretion of the Investigator, on a case by case basis, changes to the regimen that might be clinically warranted may be made prior to Week 24 after consulting with the Medical Monitor and obtaining approval.

Sites are required to indicate if a medication is used for prophylaxis purposes or if it is used for the acute treatment of migraines. The Investigator should reevaluate the patient's risk factors relative to the prescribing information for both prophylactic and acute treatments that the patient is using, and judge that the use of these medications continues to be considered safe.

# 10. STUDY ASSESSMENTS AND PROCEDURES

# **10.1.** Schedule of Assessments

Assessment and procedures at each visit are summarized in Section 2 - Schedule of Events and Assessments.

# 10.2. Assessments and Procedures

# 10.2.1. Randomization

Randomization must occur after the subject completes the 28-day eDiary screening period. Every effort should be made to conduct an onsite randomization visit; however, a phone visit is acceptable in cases where the subject's schedule will not permit an onsite visit.

All subjects will be randomized via the IWRS (Interactive Web Response System) after the following:

- Eligibility has been approved by the Medical Monitor
- Review of all inclusion/exclusion criteria to confirm subject continues to meet inclusion/exclusion criteria.
- Verification that subject meets eDiary-related eligibility criteria as calculated within the eDiary portal.
- Subject confirms continued interest in participating in the study.

# 10.2.2. Demographics

The year of birth, age, sex, ethnicity, race, and how the subject was recruited to the study will be collected in source records and in the CRF.

# **10.2.3.** Medical History

Significant historic and current medical conditions or illnesses, allergies to medications, and prior surgical interventions will be recorded in the source records and in the CRF. Symptoms that are ongoing at the time of informed consent will be considered medical history.

Migraine history will also be collected in the source records and the CRF, including age at diagnosis of chronic migraine as well as other details of the subjects' history with migraine. If

the subject is not a current or past user of a prescribed or over-the-counter medication for migraine, the Medical Monitor will be consulted.

Investigators should demonstrate due diligence in trying to obtain medical records. All attempts to obtain medical records should be documented. If medical records cannot be obtained, history may be confirmed via patient interview in order to obtain sufficient information to confirm all eligibility criteria are met.

# 10.2.4. Physical Examinations

Physical examinations will be performed at the times noted in the Schedule of Events and Assessments in Section 2 and must be performed by an Investigator who has been trained and delegated the task on the Delegation of Authority Log.

The physical examination at the screening visit will be comprehensive and appropriate to determine the overall physical health of each subject. Examination of the genitourinary system and rectum may be deferred by the Investigator if the subject's related medical history and review of systems are negative. For all other visits that call for a physical examination, the body systems examined will be at the discretion of the Investigator.

Each physical examination will include weight measurement. Height will be measured at screening only.

Abnormal physical examination findings at the screening visit will be recorded as medical history. Any new or worsening physical examination finding identified after informed consent will be considered an AE.

# **10.2.5.** Vital Signs

Vital signs, including blood pressure (BP) and pulse, will be measured at the time points specified in the Schedule of Events and Assessments in Section 2.

When measuring vital signs, the subject should be seated comfortably, with back supported and rested for 5 minutes before obtaining vital signs. Blood pressure may be repeated to confirm measurement.

For BP measurements, the subject should have their upper arm positioned so that it is level with their heart and feet flat on the floor. Excess clothing that might interfere with the BP cuff or constrict blood flow in the arm should be removed. A blood pressure cuff of appropriate size should be wrapped around the bare upper arm such that the bladder portion of the cuff extends at least 80% around the arm. The center of the bladder should be in line with the brachial artery so as to allow the stethoscope diaphragm clear access to the brachial artery. Site staff and subject should refrain from talking during the reading.

# 10.2.6. **Questionnaires**

Questionnaires should be administered to subjects in the order listed below. On Day 0 and Week 12, all questionnaires should be administered prior to dosing.

Protocol number, subject number and date of administration must be captured on all questionnaires. All questionnaires completed by subjects must be reviewed for completeness and clarity by site staff prior to the subject leaving the clinic. The subject should be asked to complete any unanswered questions.

# 10.2.7. Columbia-Suicide Severity Rating Scale (C-SSRS)

The C-SSRS will be administered by trained (i.e., C-SSRS certified) site staff at the time points specified in the Schedule of Events and Assessments in Section 2. The C-SSRS must be administered prior to dosing at dosing visits (Day 0 and Week 12).

The C-SSRS "Baseline/Screening" version will be used for the Screening Visit, and the C-SSRS "Since Last Visit" version will be used for all subsequent visits.

# 10.2.8. Most Bothersome Symptom (MBS)

The Investigator will verbally obtain the most bothersome symptom associated with the subject's migraines during the screening visit. The most bothersome symptom will be captured in the eCRF and may include nausea, vomiting, sensitivity to light, sensitivity to sound, mental cloudiness, fatigue, pain with activity, mood changes, or other migraine-related symptom.

At each subsequent visit, the site staff will provide the questionnaire along with the other subject-completed questionnaires as specified in the Schedule of Events and Assessments in Section 2.

### 10.2.9. Other Ouestionnaires

The following questionnaires will be administered at days and times provided in the Schedule of Events in Section 2. Subjects will be given the questionnaires in the order specified below and asked to review the brief instructions on each questionnaire and complete.

- Patient Global Impression of Change (PGIC)
- Short-Form Health Survey (SF-36)
- Health-Related Quality of Life (EQ-5D-5L)
- Headache Impact Test (HIT-6)

### 10.2.10. 12-Lead ECG

ECGs will be performed using a 12-lead ECG device provided for the study at the time points specified in the Schedule of Events and Assessments in Section 2. On Day 0 and at Week 12, ECG must be performed pre-dose, and within 2 hours post-dose. ECG data will be transmitted and read centrally by a cardiologist; however, the Investigator must review the ECG prior to dosing and ensure there are no clinically significant abnormalities prior to dosing. In addition, all confirmed (i.e., centrally-read) ECGs will be reviewed by the Investigator and evaluated for clinical significance in a timely manner.

All ECGs are expected to be performed on the ECG device provided to the site by the trial Sponsor. A local ECG device may be used only in the event that there are technical issues with the central ECG device that cannot be resolved while the subject is onsite. If a local ECG device is used, a paper ECG must be submitted to the ECG vendor for central reading. All technical issues must be reported immediately to the ECG vendor help desk.

# 10.2.11. Laboratory Samples and Testing

# 10.2.11.1. Urine Drug Screening

Drugs of abuse screening test will be performed on urine samples during the screening visit. Urine drug screen kits will be provided by the central lab and the test performed on site. If a urine drug screen is positive and there is no medical record documentation of prescribed medications to explain the result, the subject should be considered for exclusion from the study. Questions regarding the eligibility can be addressed with the Medical Monitor.

# 10.2.11.2. Pregnancy Testing

Urine pregnancy tests will be performed for all female subjects, regardless of childbearing potential, at the specified time points in the Schedule of Assessments, Section 2. On Day 0 and at Week 12, urine pregnancy test must be performed prior to dosing.

Urine pregnancy test kits will be provided by the central lab, and the test performed on site.

The contraceptive method used by females of child-bearing potential and males with partners of child-bearing potential must be confirmed with the subject and recorded in the source record at screening, and reconfirmed with the subject and recorded in the source record at each subsequent study visit.

# 10.2.11.3. Clinical Laboratory Testing

Blood samples for clinical laboratory tests, including hematology, serum chemistry and serology (including HIV, Hepatitis B and Hepatitis C), will be collected at the time points specified in the Schedule of Events and Assessments in Section 2. Clinical laboratory tests performed are listed in Section 11.1.7.

All clinical laboratory blood samples will be initially processed by site staff and shipped to a central laboratory for analysis as specified in the Laboratory Manual. An Investigator listed on the Form FDA 1572 will review all lab reports and document clinical significance for any out-of-range lab value(s) listed in the report.

# 10.2.11.4. Pharmacokinetic and Immunogenicity Sampling

Blood samples will be collected for the analysis of plasma PK of ALD403 and for determination of anti-ALD403 antibodies in serum (immunogenicity) at specified time points in the Schedule of Events and Assessment in Section 2. All samples will be initially processed, stored, and shipped as specified in the Laboratory Manual.

# 10.3. eDiary Completion and Compliance Review

The subject will be instructed to complete an electronic diary (eDiary) daily from screening through Week 24.

The eDiary will be distributed to each subject at the screening visit after subject training on eDiary use by site staff. The day of eDiary distribution will start the 28 day eDiary screening

period. The subject will record information daily regarding headache characteristics, severity, and length. During the screening period, an eDiary Eligibility Report will summarize baseline headache and migraine days and eDiary compliance. The headache and compliance data from the eDiary will also be made available to the clinical site for review on a regular basis via the eDiary system portal.

Subject eligibility will be confirmed prior to randomization. Any subject found to be ineligible for the study during the screening period or prior to randomization or dosing will not be randomized or dosed.

Site staff will monitor each subjects eDiary compliance on an ongoing basis through Week 24, and will counsel subjects as needed on the on the importance of completing the eDiary daily. All follow-up with subjects regarding eDiary compliance should be documented in the source records.

During the Week 24 visit, or Early Termination visit if subject discontinues prior to Week 24, eDiary closeout must be performed while the subject is on site.

# 11. ASSESSMENT OF SAFETY

# 11.1. Adverse Events

### 11.1.1. Definitions

An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product that does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. (ICH E6)

### 11.1.2. Assessment of Adverse Events

The Investigator is required to monitor the occurrence of adverse events for each subject from the time of informed consent through the course of the clinical trial. Adverse events may be reported by the subject, reported by a caregiver, or reported by the investigative site through Investigator site personnel open-ended questioning, through physical examination, laboratory test, documentation in medical records, or by other means. Adverse events include:

- Any new undesirable medical experience or an unfavorable and unintended change of an
  existing condition that occurs during or after treatment, whether or not considered related
  to the Investigational Product.
- Any abnormal assessment or laboratory findings considered by the Investigator to be
  clinically significant. Clinically significant findings include but are not limited to those
  that lead to discontinuation or interruption of study treatment, require therapeutic
  intervention, or require a change in subject management.

A new or worsening of a pre-existing or chronic condition is considered an adverse event and must be reported as such. Medical conditions, which existed prior to the time of informed consent into the clinical trial, will not be considered an adverse event unless the condition worsens. Unchanged, chronic, non-worsening or pre-existing conditions from the time of informed consent are not adverse events and should not be recorded on the AE eCRF.

Pre-existing medical conditions of clinical significance must be included in the subject's medical history and recorded on the medical history eCRF page.

Each event recorded on the AE eCRF is required to be assessed by the Investigator with regard to the following; seriousness, severity, and relationship to Investigational Product, as outlined below.

### Seriousness

An adverse event or suspected adverse event is considered serious if in the view of either the Investigator or Sponsor, it results in;

- Death
- Is life-threatening (this means that the subject is at risk of death at the time of the event; it does not mean that the event hypothetically might have caused death if it were more severe)
- Inpatient hospitalization or prolonged existing hospitalization
- A persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions.
- Congenital anomaly/ birth defect
- Important medical events that may not result in death, be life-threatening or require hospitalization may be considered serious when, based upon appropriate medical judgement, they may jeopardize the patient or subject and/or may require medical or surgical intervention to prevent one of the outcomes listed in the definition (21 CFR 312.32(a) and ICH E2A).

### Of note:

- A social hospitalization (i.e., hospitalizations for pre-admissions not due to an acute medical issue) is not considered an SAE
- Hospitalization is considered a greater than 24 hour hospital admission.

# **Severity**

The severity of an AE will be graded as follows:

 Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.

- Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting ageappropriate instrumental Activities of Daily Living (ADL).
- Grade 3 Severe or medically significant but not immediately life-threatening;
   hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL.
- Grade 4 Life-threatening consequences; urgent intervention indicated.
- Grade 5 Death related to AE.

# **Relationship to Investigational Product**

The Investigator is required to assess the causality/relationship between each AE and the Investigational Product as not related or related and record the assessment on the source documents and in the eCRF AE page. Medical judgment should be used to determine the likely relationship of the AE to the Investigational Product considering all relevant factors including (but not limited to) relevant history, concomitant medical condition and concomitant medications. Determination should be based on assessment of temporal relationships, biologic plausibility, association (or lack of association) with underlying disease, and presence (or absence) of a more likely cause.

**Not Related:** It is plausible that the AE has an etiology other than the Investigational Product (e.g., pre-existing condition, underlying disease, concomitant medical condition, or concomitant medication).

**Related:** The AE cannot reasonably be explained by the subject's clinical state, concomitant medical condition or concomitant therapies, and a temporal relationship exists between the event onset and administration of the Investigational Product.

# 11.1.3. Recording Adverse Events

Event reporting will extend from time of informed consent until completion of the final visit. Serious adverse events occurring after the end of the clinical trial must be reported if the Investigator considers there to be a causal relationship with the Investigational Product.

SAE Notification Form should be used to report any related SAEs which occur after the end of the clinical trial.

Adverse events (AEs) should be recorded on the AE eCRF, whether believed by the Investigator to be related or not related to the Investigational Product.

AE reporting should contain:

- A brief description of the event
- Date of onset
- Date of resolution
- Severity
- Actions taken or treatment required
- Relationship to Investigational Product
- Outcome
- Whether the event is considered serious

Whenever possible, the Investigator should group signs or symptoms that constitute a single diagnosis into a single event term. For example, "cough, rhinitis, and sneezing" might be grouped together as "upper respiratory tract infection."

Asymptomatic abnormal findings considered by the Investigator to be clinically significant should be recorded as an AE, unless it is associated with a clinical syndrome that has already been reported as an AE.

# 11.1.4. Reporting Serious Adverse Events

All SAEs that occur during the period of observation, whether considered to be related to the Investigational Product or not, must be reported within 24 hours of awareness or knowledge of the event. The date the site personnel became aware of the serious adverse event must be recorded in the source document. To report the SAE, complete the eCRF AE page and indicate the reason for seriousness. The minimum information required for an initial report is:

- Sender of report (name, address of Investigator)
- Subject identification (screening/randomization number, initials, NOT subject name)
- Protocol number

- Description of SAE (e.g., event term)
- Seriousness criteria
- Relationship assessment

After receipt of the initial report, the Medical Monitor or designee will review the information and, if necessary, contact the Investigator to obtain further information for assessment of the event. The Sponsor or designee will be responsible for information processing and reporting in accordance with applicable local and regulatory requirements.

The Sponsor will determine if an SAE requires expedited reporting to regulatory agencies. The clinical trial site personnel are responsible for reporting these events to their EC/IRB according to the institution's EC/IRB reporting requirements and in accordance with applicable local and regulatory requirements.

Should the EDC System not be available, serious adverse events must be reported on the paper SAE Notification Form. Additional details can be found in the Site Manual. This does not replace the EDC reporting system; information must be entered in the EDC system once the system returns to normal function.

# 11.1.5. Unexpected and Related Serious Adverse Events

Unexpected SAEs are those which:

- Are not previously reported as associated with ALD403, as referenced in the Investigator's Brochure.
- May be symptomatically and pathophysiologically related to an AE listed in the Investigator's Brochure, but differ from the event due to greater severity, frequency or specificity.

The Sponsor or designee will report, to the appropriate regulatory authorities according to local and regulatory requirements, unexpected SAEs which are considered related to ALD403 (suspected unexpected serious adverse reactions [SUSARs]). The clinical trial site personnel are responsible for reporting these events to their EC/IRB in accordance with applicable local and regulatory requirements.

# 11.1.6. Follow-up of Adverse Events

Irrespective of the suspected causality, AEs will be monitored until resolution, stabilization in the judgment of the Investigator, or the subject is lost to follow up or withdraws from the trial.

# 11.1.7. Clinical Laboratory Tests

Serum chemistry tests include albumin, alkaline phosphatase (ALP), alanine aminotransferase (ALT), aspartate aminotransferase (AST), urea nitrogen, calcium, bicarbonate, creatinine, globulin, glucose, phosphorus, potassium, sodium, total bilirubin, total cholesterol, total protein, triglycerides, magnesium and uric acid.

Hematology tests include hematocrit, hemoglobin, platelet count, red blood cell (RBC) count, and white blood cell (WBC) count with differentials (neutrophils, lymphocytes, monocytes, eosinophils, and basophils).

# 11.1.8. Pregnancy

In the event that a female subject becomes pregnant following administration of Investigational Product or may have been pregnant at the time of Investigational Product exposure, or the partner of a male subject becomes pregnant following administration of Investigational Product, the pregnancy must be reported to the Sponsor within five business days of the Investigator becoming aware of the pregnancy. Pregnancy information will be reported to the Sponsor using the Exposure In-Utero Forms in EDC. An Exposure In-Utero Notification Form should be used to report a pregnancy that occurs within 30 days after study completion of the trial.

Although pregnancy *per se* is not considered an AE, the outcome of a pregnancy that results in a birth defect or congenital anomaly or hospitalization for any reason is considered to be an SAE. Every attempt should be made to follow a pregnancy to conclusion.

Follow-up information is to be collected by the Investigator and provided to the Sponsor regarding:

- The course of the pregnancy including perinatal and neonatal outcome, premature termination of the pregnancy, or miscarriage
- Offspring information including birth weight and birth defects (if any)

### 11.1.9. Suicidal Ideation and Behavior

Recent meta-analyses, spontaneous reports, and published case reports regarding suicidal ideation and behavior arising from drugs tested in clinical trials have been noted as an area of general concern. Based on this information, the United States Food and Drug Administration (FDA) has provided guidance to prospectively assess suicidal ideation and behavior in clinical trials to ensure that subjects in clinical trials who are experiencing suicidal ideation and behavior are properly recognized and adequately treated and to ensure the collection of more timely and more complete data on suicidal ideation and behavior than have been collected in the past. The C-SSRS (Columbia-Suicide Severity Rating Scale) will be used for this purpose. Any subject who answers "yes" to questions 4 or 5 of the C-SSRS during the screening visit will be referred to a mental health specialist by the Investigator. During the course of the trial after dosing, any subject who answers "yes" to questions 4 or 5 of the Suicidal Ideation section or answers "yes" to any question in the Suicidal Behavior section of the C-SSRS will be discontinued from the study treatment as specified in Section 8.4.1, and referred by Investigators to a mental health specialist. Affirmative answers to questions 4 or 5 for suicidal ideation or to any question for suicidal behavior will be reported in EDC as an AE.

# 11.2. Management of Reactions to ALD403

There are no specific antidotes to ALD403.

Each medical emergency should be treated appropriately by the Investigator using proper standard of care, according to their typical clinical practice and local guidelines for that emergency condition. Emergency equipment and medication for the treatment of these potential adverse events must be available for immediate use.

Should a medical condition arise that the Investigator believes is related to the Investigational Product, clinical judgment should be used to provide the appropriate response including the consideration of discontinuation of Investigational Product. Any events believed to be potential allergic reactions should be discussed with the Medical Monitor.

If a subject experiences a potential systemic allergic reaction, as assessed by the Investigator, the site will collect additional blood specimens using the immune response lab kit, per the laboratory manual, at the time of the event and again at the next scheduled visit. This assessment includes serum histamine, serum tryptase, immunoglobulin E, and complement components. Subjects

who have experienced a potential significant allergic reaction after administration of Investigational Product should not receive subsequent doses.

Whether maintained in a "formal crash cart" or separately, the following is a requirement at the site:

- CPR certification by site staff performing study assessments
- Automated external defibrillator (AED)
- Emergency medications including antihistamines, bronchodilators, IV saline, corticosteroids, acetaminophen, and epinephrine

The AED and emergency medication should be immediately available on an Investigational product infusion day.

# 12. ASSESSMENT OF EFFICACY, PHARMACOKINETICS, AND IMMUNOGENICITY

# 12.1. Efficacy

# **12.1.1. eDiary**

Subjects will complete a daily headache eDiary from the time of screening to Week 24. The eDiary should be completed each trial day whether or not the subject had a headache. These daily entries record if the subject took acute migraine medication on that day. The eDiary data from the 28 days following screening visit will be used to determine eligibility criteria, and the baseline migraine and headache results.

# 12.1.2. Endpoints

Headache episodes will be self-reported by the subject. An episode is a single headache event that the subject reported as having a start and an end and which lasts at least 30 minutes. The term headache will encompass both headaches and migraine headaches. The migraine and headache endpoints will be summarized in 4-week intervals. Specifically, migraine and headache endpoints will be summarized for the 4-week intervals: Weeks 1-4, 5-8, 9-12,...21-24, the 12-week intervals: Weeks 1-12, 13-24, and the 24-week interval: Weeks 1-24.

### Migraine Day

A migraine day is defined as any day with a headache that meets the chronic migraine definition as outlined in the International Headache Society (IHS) International Classification of Headache Disorders (ICHD, 3<sup>rd</sup> edition, beta version 2013), Section 1.3 with diagnostic criteria C limited to items 1 and 3.<sup>4</sup> Criteria C defines what characteristics must be present for a headache to be considered a migraine. These characteristics define a migraine as a self-reported headache that:

### 1. Lasted

- a. 4 hours or more or
- b. 30 minutes to 4 hours, and believed by the subject to be a migraine that was relieved by medication
- 2. Had at least 2 of the following:
  - a. Unilateral location
  - b. Pulsating quality

- c. Moderate or severe pain intensity
- d. Aggravation by or causing avoidance of routine physical activity
- 3. Had at least 1 of the following:
  - a. Nausea and/or vomiting
  - b. Photophobia and phonophobia

Frequency, Change and Percent Change of Migraine Days/Headache Days

The frequency of migraine days is the number of migraine days within four week intervals and the average four week frequency in twelve and twenty-four week intervals. Change from baseline is the difference in frequency between baseline and the counts within these four week intervals. The 12 and 24 week change is the difference in the frequency between baseline and the average of the, 4 week intervals. The percent change is 100 times the ratio of the change and the baseline frequency. Similar measures will be produced based upon headache frequency.

# Migraine/Headache Responder Rate

Three responder rates will be utilized: 50%, 75% and 100%. A responder is a subject who achieves a  $\geq$ 50% reduction,  $\geq$ 75% reduction, or 100% reduction in migraine days, respectively. These reductions will be evaluated by comparing the baseline frequency of migraine days to the migraine frequency in four week intervals. The same analyses will be conducted for headache days.

Results from these four week intervals will be combined to produce 12 and 24 week responder endpoints. The Weeks 1-4, 5-8, and 9-12 change from baseline measures are averaged, and the average value is compared to baseline. A percent change from baseline is determined, which is used to determine the responder status. A 75% migraine responder will be a subject who achieves the specified percent reduction in migraine days within these intervals based upon the average change from baseline measures. A 50% migraine responder will be similarly defined.

A 100% migraine responder rate over Weeks 1-12, 13-24 and 1-24 is the average of the 100% responder rate for four week intervals that make up these intervals. Hence, the 100% migraine responder rate over weeks 1-12 is the average of the 100% migraine responder rates in Weeks 1-4, 5-8 and 9-12 for the treatment arm.

Time to First Migraine

Time to the first migraine after dosing will be analyzed based upon the migraine data entered into the eDiary.

Migraine Hours/Headache Hours

Migraine hours are the sum of the duration of migraines within four week intervals, and the average four week duration within 12 and 24 week intervals. Headache hours are similarly defined but include all headaches. Subjects with no migraines/headaches will have a duration of zero.

Acute Medication Usage

The percent of migraines and headaches with acute medication use will be summarized. Subjects with no migraines/headaches will be included with a rate of zero.

Acute Migraine Medication Usage

The number of days that subjects used acute migraine medication (i.e. triptan or ergotamine) will be summarized in 4, 12, and 24 week intervals. The 12 and 24 week results will be the average of the individual 4 week results that make up those wider intervals (e.g. the secondary endpoint of Weeks 1-12 will be the average of the Weeks 1-4, 5-8, and 9-12 results). The change from baseline for these measures will be the difference between the post baseline interval and baseline.

Percentage of subjects with a migraine on the day after dosing

The percent of subjects with a migraine on the day after dosing will be summarized Reduction in migraine prevalence from baseline to Week 4

The average percent of subjects with a migraine on any given day during baseline and the equivalent average rate over Weeks 1, 2, 3 and 4 will be evaluated for the active and the control arms.

Migraine/Headache Severity

Headache severity will be collected on a 3 point scale: mild pain, moderate pain, severe pain. Subjects with no migraines/headaches will be concerned as having zero percent of severe pain migraines/headaches.

Patient Global Impression of Change (PGIC)

The PGIC includes a single question concerning the subject's impression of the change in their disease status since the start of the study. Seven responses are possible: Very Much Improved, Much Improved, Minimally Improved, No Change, Minimally Worse, Much Worse, Very Much Worse.

SF-36 Health Survey (SF-36 v2.0)

The SF-36 v2.0 is a health survey containing 36 questions consisting of eight scaled scores to measure quality of life over the past 4 weeks, see Appendix 15.3. The eight sections measured are vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health. These sections are combined into the mental component score and physical component score.

*EQ-5D-5L* 

The EQ-5D-5L is a descriptive system of health-related quality of life states consisting of five dimensions/questions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each of which can take one of five responses. The responses record five levels of severity (no problems/slight problems/moderate problems/severe problems/extreme problems) within a particular EQ-5D dimension. The EQ-5D-5L additionally includes a VAS scale. Each item will be summarized separately.

Headache Impact Test (HIT-6 v1.0)

The Headache Impact Test (HIT) is a tool used to measure the impact and effect on the ability to function normal in daily life when a headache occurs. The HIT is a 6 question, Likert-type, self-reporting questionnaire with responses ranging from "Never" to "Always" with the following response scores: Never=6, Rarely=8, Sometimes=10, Very Often=11, Always=13. See Appendix 15.3. The total score for the HIT is the sum of each response score and will be treated as missing if the response is missing for one or more questions. The HIT total score ranges from 36 to 78, with score ranges having the following life impact:

| Score Range | Life Impact |
|-------------|----------------|
| >= 60 | Severe |
| 56-59 | Substantial |
| 50-55 | Some |
| <= 49 | Little to None |

Migraine Attack/Headache Episode

A migraine attack is defined as 1 continuously recorded migraine. One attack may result in multiple migraine days. Headache episodes are similarly defined.

Migraine symptom-free days

The number of days the subject is free of migraine symptoms (e.g. pulsating, moderate or severe pain, nausea) will be summarized for each 4-week period.

Most Bothersome Symptom (MBS)

At screening subjects will identify migraine related symptom that is most bothersome for them. Subjects will be asked to rate the improvement in this symptom from screening on a seven-point scale identical to the scale used for the PGIC.

# 12.2. Pharmacokinetics

The concentrations of ALD403 will be measured in plasma from all ALD403-treated subjects using a validated assay. The PK analysis will include evaluations of concentration-time profiles for free ALD403 at the following times: pre-dose on Day 0, immediately post-dose (within 15 minutes of end of infusion) and Weeks 2, 4, 8, 12 (pre-dose), 24, and 32 or ET.

For subjects receiving placebo, selected plasma samples may be analysed for the potential presence of ALD403 using a validated assay.

All plasma PK samples will be stored at -20°C or below prior to shipping to the central laboratory.

Additional sample handling, processing, storage, labelling and shipping instructions will be provided to the site in a laboratory manual.

If a subject terminates early from the clinical trial, all efforts will be made to collect blood samples to analyse for free ALD403 unless consent has been withdrawn.

# 12.3. Immunogenicity

Serum blood samples will be taken pre-dose on Day 0, and Weeks 2, 4, 8, 12 (pre-dose), 24, and 32 or ET to test for the development of antibodies to ALD403. The immunogenicity will be

assessed in serum from all ALD403-treated subjects using a validated assay. Immunogenicity will not be assessed in placebo subjects.

If a subject terminates early from the clinical trial, all efforts will be made to collect blood samples to analyze for antibodies against ALD403 unless consent has been withdrawn. For any samples that are positive for anti-ALD403 antibody, there may be additional testing to characterize the anti-ALD403 antibody for the potential to neutralize (NAb) ALD403 activity. Subjects who test positive for specific anti-ALD403 antibodies at the time of the last study visit will be asked to provide up to 2 additional blood samples for immunogenicity testing at 3 month intervals for up to 6 months.

Additional sample handling, processing, storage, labelling and shipping instructions will be provided to the site in a laboratory manual.

# 13. STATISTICAL CONSIDERATIONS

# 13.1. Decision Rule

A multiplicity procedure will be used to account for multiplicity of dose levels for the primary endpoint and the key secondary endpoints. This procedure will start with the 300 mg vs placebo comparison for the primary endpoint. If this is significant, testing will continue to key secondary endpoints for 300 mg. The procedure will then move on to the 100 mg group for the primary endpoint and subsequently the secondary endpoints. Statistical testing will be conducted to maintain study wide two-sided 5% alpha level.

# 13.2. Sample Size

The planned sample size for this study is 1050 randomized and treated subjects. These subjects will be allocated into 3 treatment groups in a 1:1:1 ratio. Pair-wise testing of each ALD403 group vs. placebo will be performed. Three hundred and fifty subjects per group provides at least 90% power for the primary endpoint for each comparison assuming a treatment effect of at least 1 day and a common standard deviation of 4 days or less. For the key secondary 75% responder rate endpoints 90% power is achieved for the pair-wise comparisons, assuming a placebo responder rate of 20%, and an ALD403 rate of 31%. These sample size calculations have been performed using Pass 2008 and are based upon a t-test and chi-squared test that should approximate the ANCOVA and CMH tests. <sup>14</sup>

### 13.3. General Considerations

### 13.3.1. Definition of Baseline

Baseline for migraine and headache endpoints will be based upon the data recorded in the headache eDiary during the 28-days following screening. For other variables, the baseline assessment will be the latest available valid measurement taken prior to the administration of Investigational Product. This will generally be Day 0.

### 13.3.2. Handling of Missing Data

Summary statistics will be reported based upon observed data except for the eDiary data which will utilize the imputation outlined below. Additionally, if the start date of an AE or concomitant medication is incomplete or missing, it will be assumed to have occurred on or after the intake of

trial medication, except if an incomplete date (e.g., month and year) clearly indicates that the event started prior to treatment.

Subjects who do not complete the eDiary daily will have missing data. It is expected that most missing eDiary data will be sporadic. If the eDiary has been completed at least 21 days in a 28 day interval, then normalization will be used. The results will be normalized to 28 days by multiplying the observed results by the inverse of the completion rate (i.e. if a subject does not complete the eDiary on 5 days they will have completed the eDiary on 82% of the days and the normalized results will be the observed results times 1.22). If the eDiary has been completed on less than 21 days in the 28 day interval then the results for the 28 day interval will be a weighted function of the observed data for the current four week interval and the results from the previous interval. The weights will be proportional to how many days the eDiary was completed and will provide greater weight to the results from the current interval as the eDiary completion rate increases. Specifically, the results will be derived as

$$28(WX_c + (1 - W)X_p),$$

where W is the days the eDiary was completed/20,  $X_c$  is the available average daily results for the current interval and  $X_p$  are the average daily results for the previous interval.

### 13.3.3. Populations to be Analyzed

The populations to be analyzed are as follows:

Full Analysis Population: Randomized subjects who received Investigational Product/placebo. Subjects will be summarized within the treatment group to which they were randomized. This population will be used for efficacy analyses.

Safety Population: Includes all subjects who received at least one dose of Investigational Product/placebo. Subjects will be summarized within the treatment group for which they actually received treatment. This population will be used for the safety analyses.

# 13.4. Statistical Methods

Continuous variables will be summarized with mean, median, standard deviation, minimum, and maximum. Categorical variables will be summarized with frequency and percentage.

# 13.4.1. Subject Disposition, Demographics and Baseline Characteristics

An accounting of all randomized trial subjects by disposition will be presented. This summarization will include a summary of all subjects who have received trial drug. Demographic, baseline characteristics, migraine history and concomitant medications (coded by the World Health Organization Drug Dictionary) will be summarized descriptively by treatment group.

# 13.4.2. Efficacy Analyses

Efficacy endpoints will be summarized with descriptive statistics. The migraine and headache endpoints will be summarized by 4, 12, and 24 week intervals with the remaining endpoints being summarized by study week.

Primary Efficacy Analyses

Hypothesis testing will be performed for the primary endpoint: change in frequency of migraine days (Weeks 1-12). This endpoint will be calculated as outlined in Section 12.1.2 and will utilize the missing data rules provided in Section 13.3.2. Summary statistics including confidence intervals for the treatment differences will be used to summarize the results for the primary endpoint. Testing will also be employed. The hypotheses tested are

$$H_o: \Delta_{plb} = \Delta_{403}$$
  $H_a: \Delta_{plb} \neq \Delta_{403}$ 

where  $\Delta_{403}$  is the change in migraine days for subjects in the ALD403 treatment arm and  $\Delta_{plb}$  is similarly defined for the placebo subjects. The change from baseline is expected to be negative as migraines are being reduced. While the test outlined above is two sided, as is the alpha level used for this study (i.e. 5%), clinically relevant results require a larger reduction of migraines on the ALD403 arms.

An ANCOVA model will be used to test for a difference between treatment arms. This model will include the change from baseline measure as the response variable. Treatment and the stratification variables: baseline migraine days (continuous predictor) and prophylactic medication use (use vs. no use) will be the independent variables.

Secondary Efficacy Analyses

Summary statistics including confidence interval for the treatment differences will be used to summarize the results for the secondary endpoints. Testing will be used for the key secondary endpoints. A CMH test controlling for the randomization stratification factors will be used for the responder rate key secondary endpoints, and the percent of subjects with a migraine on the day after dosing endpoint will be tested with an extended CMH test.<sup>15</sup>

The acute migraine medication day endpoint will be tested using an ANCOVA model similar to the one used for the primary endpoint. The time to first migraine analysis will be descriptively summarized based upon Kaplan-Meier methods.

The missing data rules provided in Section 13.3.2 will be used for the key secondary endpoints, except for the percentage (prevalence) of subjects with a migraine on the day after dosing endpoint. Subjects who did not complete the eDiary on the day following dosing will be included in the prevalence rate calculation based upon their Week 1-4 daily migraine rate. Hence, subjects with a migraine will be included in the rate calculation as a value of 1, subjects who completed the eDiary and did not have a migraine will be included as a 0, and subjects who did not complete the eDiary will be included with a value between 0 and 1 equal to their prevalence rate in Weeks 1-4 (i.e. the number of Weeks 1-4 migraine days divided by 28). The reduction in migraine prevalence from baseline to Week 4 endpoint will be difference in daily prevalence rates between Week 1 and baseline, Week 2 and baseline, and so on. The baseline daily prevalence will be calculated as the number of migraine days in baseline divided by 28. The Week 1 daily prevalence will be the number of migraine days in Week 1 divided by 7, with a similar definition for Weeks 2, 3, and 4. The same missing data approach for the day after dosing endpoint will be used for these weekly measures (i.e. any day the subject does not complete the diary will be assigned a value equal to the Weeks 1-4 prevalence rate). The treatment effect will be evaluated using a repeated-measures approach.<sup>16</sup> The model will specify an unstructured variance/covariance matrix and include the treatment group, visit, baseline value of the outcome variable and treatment group-by-visit interaction. The Kenward-Roger approximation will be used to estimate the degrees of freedom. Pharmacokinetic Analyses

# 13.4.3. Analysis of Drug Concentrations

The concentrations of ALD403 will be listed and summarized by time point and dose group, and descriptive statistics will be provided. In this analysis, concentrations below the lower limit of quantification (LLOQ) will be set to zero.

Plots of the individual concentrations of ALD403 will be presented over time (linear and log scales). Plots of the mean or median concentration will be presented over time (linear and log scales). When the scale is linear, concentrations below the lower limit of quantification will be set to zero. In the log-scaled figures, concentrations below the LLOQ will be imputed as LLOQ/2. Population pharmacokinetic analysis will be performed on the results for ALD403 concentrations obtained during this study in combination with the results from other studies of ALD403 in normal subjects and migraine patients.

# 13.4.4. Safety Analyses

## 13.4.4.1. Adverse Events

The incidence of all AEs will be tabulated by treatment received. These AEs will be classified by system organ class and preferred term using the Medical Dictionary for Regulatory Activities (MedDRA). For incidence reporting, if a subject reported more than 1 AE that was coded to the same preferred term/system organ class, the subject will be counted only once for that specific preferred term/system organ class. Events recorded between the time the informed consent is signed and the first Investigational Product administration will be listed.

An overview of AEs, which includes subject incidence of AEs, SAEs, deaths, and AEs leading to discontinuation, will be presented. For AEs presented by severity, the worst severity during the clinical trial will be presented for each subject.

The subject incidence of AEs will be summarized by system organ class and preferred term.

### 13.4.4.2. Serious Adverse Events

All SAEs will be listed and summarized in a similar manner to AEs.

### 13.4.4.3. Clinical Laboratory Results

Summary statistics for actual values and for changes from baseline will be tabulated for clinical laboratory results by scheduled visit. Subjects with clinical laboratory values outside of the

normal reference range at any post-baseline assessment will be summarized. Shifts from baseline clinical laboratory values based upon the normal range and will be tabulated. Subjects developing an antibody response will be listed.

# 13.4.4.4. Electrocardiogram (ECG) Results

The observed data at baseline and change from baseline for each measurement day will be summarized with descriptive statistics.

# **13.4.4.5.** Vital Signs

The observed data at baseline and change from baseline for each measurement day will be summarized with descriptive statistics.

### 13.4.4.6. C-SSRS

The C-SSRS assesses lifetime suicidality during an initial baseline evaluation, and then monitors suicidal ideation and suicidal behavior at subsequent follow-up assessments. Four constructs are measured. The first and second are the severity and intensity of ideation, rated on a 5-point ordinal scale. The third is the behavior subscale, which is rated on a nominal scale and the fourth is the lethality subscale, which assesses actual attempts. These results will be reported at baseline and post baseline. Results for individual time points will be provided in a listing.

# 14. ETHICAL, LEGAL AND ADMINISTRATIVE ASPECTS

# **14.1.** Data Quality Assurance

The Sponsor or designee will assess the site to verify the qualifications of each Investigator, according to Sponsor's or applicable SOPs. There will be an inspection of site facilities, and Investigator will be further informed of responsibilities and the procedures for ensuring adequate and correct documentation.

The Investigator is required to prepare and maintain adequate and accurate case histories designed to record all observations and other data pertinent to the clinical trial for each clinical trial subject. All information recorded on the CRFs for this clinical trial must be consistent with the subjects' source documentation (i.e., medical records).

# 14.2. Case Report Forms and Source Documents

As part of the responsibilities assumed by participating in the study, the principal investigator or sub-investigator agrees to maintain adequate case histories for the patients treated as part of the research under this protocol. The principal investigator or sub-investigator agrees to maintain accurate eCRFs and source documentation as part of the case histories. These source documents include, but are not limited to, laboratory reports and original ECGs.

# 14.3. Study Documentation

Source document is defined as any hand written or computer generated document that contains medical information or test results that have been collected for or are in support of the protocol specifications, e.g., clinical laboratory reports, clinic notes, drug disbursement log, subject sign in sheets, subject completed questionnaires if applicable, telephone logs, ECGs, etc. All draft, preliminary and pre-final iterations of a final report are also considered to be source documents, e.g., faxed laboratory reports and hard copy laboratory reports, faxed initial results and hard copy, final report.

# 14.4. Data Collection and Electronic Data Capture (EDC)

The data collected during the study (except clinical laboratory test results, eDiary results, ECG results, PK analyses, Immunogenicity) will be recorded in the subject's eCRF. The Short-Form Health Survey (SF-36), Health related Quality of Life (EQ-5D-5L), Headache Impact Test (HIT-

6), Patient Global Impression of Change (PGIC), Most Bothersome Symptom (MBS) and C-SSRS will be completed on paper forms and then entered into the EDC system. The study site(s) will use an EDC system that is compliant with relevant Food and Drug Administration (FDA) regulatory requirements per 21 CFR Part 11. Data queries and data corrections will be handled through the same system. All transactions within the EDC system are fully documented within an electronic audit trail. Each set of completed eCRFs must be reviewed after being source verified by monitor and electronically signed and dated by the Investigator.

# 14.5. Archiving Clinical Trial Records

According to ICH guidelines, essential documents should be retained for a minimum of 2 years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or at least 2 years have elapsed since the formal discontinuation of clinical development of the Investigational Product. However, these documents should be retained for a longer period if required by applicable legal requirements.

It is the responsibility of the Investigator and clinical trial staff to maintain a comprehensive and centralized filing system of all clinical trial-related documentation. This centralized file should be available for inspection at any time by the Monitor or Quality Assurance staff for monitoring or auditing by Alder BioPharmaceuticals, Inc. and regulatory authorities. Elements of clinical trial documentation should include:

- Subject files containing the completed CRFs supporting source documentation and the signed ICF
- Clinical trial files, containing the protocol with all amendments, the Investigator
  Brochure, copies of all clinical trial documentation, and all correspondence to and
  from the ethics committee and Alder BioPharmaceuticals, Inc.
- Pharmacy files, containing the Investigational Product Accountability Records or dispensation logs and all clinical trial agent-related correspondence

# 14.6. Good Clinical Practice

The procedures set out in this clinical trial protocol are designed to ensure that the Sponsor and Investigator abide by the principles of the GCP guidelines of the ICH and applicable federal and

local regulations. The clinical trial also will be conducted in keeping with local legal requirements.

# 14.7. Informed Consent

Before each subject is admitted to the clinical trial, informed consent will be obtained from the subject (or his/her legally authorized representative) according to the regulatory and legal requirements of the participating country. The consent forms must be dated and retained by the Investigator as part of the clinical trial records. The Investigator will not undertake any investigation specifically required for the clinical trial until valid consent has been obtained. The terms of the consent and when it was obtained must also be documented in the CRF. Each subject will receive a fully-signed copy of each consent form that he/she signs for the clinical trial.

If a protocol amendment is required, the ICF may need to be revised to reflect the changes to the protocol. If the consent form is revised, it must be reviewed and approved by the appropriate ethics committee, and signed by all subjects subsequently enrolled in the clinical trial as well as those currently enrolled in the clinical trial. If subject or subject's partner, becomes pregnant during their participation in the trial, a separate pregnancy informed consent form will be obtained, to follow the pregnancy, any complications, and the health of the baby. The pregnancy consent should be obtained at the time the Investigator becomes aware of the pregnancy.

# 14.8. Protocol Approval and Amendment

Before the start of the clinical trial, the clinical trial protocol and/or other relevant documents will be approved by the ethics committee, in accordance with local legal requirements. The Sponsor must ensure that all ethical and legal requirements have been met before the first subject is enrolled in the clinical trial.

The procedures outlined in the protocol and eCRFs will be carefully reviewed by the Investigator and staff prior to clinical trial initiation to ensure appropriate interpretation and implementation. No deviations from the protocol should be made except in emergency situations where alternative treatment is necessary for the protection, proper care and well-being of subjects.

This protocol is to be followed exactly. To alter the protocol, amendments must be written, and approvals must be received from the appropriate personnel and from the ethics committee before

implementation (if appropriate). Amendments will originate from Alder BioPharmaceuticals, Inc., and will be provided to the Investigator for submission to his/her ethics committee for their review and approval prior to implementation (if appropriate). It should be noted that when an amendment to a protocol substantially alters the clinical trial design or increases potential risk to the clinical trial subject, the ICF should be revised and, if applicable, subject's consent to continue participation should be obtained.

Administrative changes may be made without the need for a formal amendment. All amendments will be distributed to all protocol recipients, with appropriate instructions.

# 14.8.1. Premature Termination of the Clinical Trial

Alder BioPharmaceuticals, Inc., reserves the right to terminate this clinical trial at any time. The FDA or other governing national authority may also terminate the clinical trial.

The Principal Investigator may discontinue participation in the trial. If the clinical trial is terminated prior to scheduled completion, the Investigator will be notified and given any necessary instructions concerning final examinations that are required. If the Investigator, the Sponsor, or the Medical Monitor becomes aware of conditions or events that suggest a possible hazard to subjects if the clinical trial continues, the clinical trial may be terminated after appropriate consultation between the relevant parties.

# 14.9. Confidentiality

All clinical trial findings and documents will be regarded as confidential. The Investigator and members of his/her research team must not disclose such information without prior written approval from the Sponsor.

The anonymity of participating subjects must be maintained. Subjects will be identified on CRFs and other documents by their subject number, initials and/or birth date, not by name and in accordance with local requirements. Documents not to be submitted that identify the subject (e.g., the signed informed consent) must be maintained in confidence by the Investigator.

# 14.10. Publication Policy

By signing the clinical trial protocol, the Investigator agrees with the use of results of the clinical trial for the purposes of national and international registration, publication, and information for

medical and pharmaceutical professionals. If necessary, the authorities will be notified of the Investigator's name, address, qualifications, and extent of involvement.

An Investigator shall not publish any data (poster, abstract, paper, etc.) without having consulted with the Sponsor in advance. The information provided in support of or generated as a result of this clinical trial is confidential. Any use or reproduction thereof, including but not limited to publications or presentations by the Investigator or his/her associates, must be submitted to Alder BioPharmaceuticals, Inc., for review and approval in accordance with the provisions contained in the clinical trial agreement. All publications must acknowledge the Sponsorship of Alder BioPharmaceuticals, Inc.

All information not previously published concerning ALD403 and Alder BioPharmaceuticals, Inc., operations, including but not limited to patent applications, formulas, manufacturing processes, basic scientific data, and formulation information, supplied by Alder BioPharmaceuticals, Inc., to the Investigator is considered confidential and shall remain the sole property of Alder BioPharmaceuticals, Inc. The Investigator agrees to use and maintain the confidentiality of this information in accordance with the provisions contained in the clinical trial agreement.

# 15. APPENDICES

# 15.1. Migraine preventive therapies with established or probable efficacy<sup>17,18,19</sup>

- Divalproex sodium
- Valproic Acid
- Topiramate
- Amitriptyline
- Venlafaxine
- Flunarizine
- Cinnarizine
- Fluoxetine
- Gabapentin
- Verapamil
- Lamotrigene
- Metoprolol
- Propranolol
- Timolol
- Atenolol
- Nadolol
- Bisoprolol
- Butterbur
- Feverfew
- Pizotifen
- Frovatriptan\*
- Naratriptan\*
- Zolmitriptan\*

Other drugs for prophylaxis will be considered on a case by case basis

<sup>\*</sup>only considered prophylaxis when specifically used as such (e.g., menstrually-related migraine (MRM))

# 15.2. Columbia-Suicide Severity Rating Scale (C-SSRS) Risk Assessment

# 15.2.1. Baseline/Screening Version

# COLUMBIA-SUICIDE SEVERITY RATING SCALE (C-SSRS)

Baseline/Screening Version

Version 1/14/09

Posner, K.; Brent, D.; Lucas, C.; Gould, M.; Stanley, B.; Brown, G.; Fisher, P.; Zelazny, J.; Burke, A.; Oquendo, M.; Mann, J.

### Disclaimer:

This scale is intended to be used by individuals who have received training in its administration. The questions contained in the Columbia-Suicide Severity Rating Scale are suggested probes. Ultimately, the determination of the presence of suicidal ideation or behavior depends on the judgment of the individual administering the scale.

Definitions of behavioral suicidal events in this scale are based on those used in <u>The Columbia Suicide History Form</u>, developed by John Mann, MD and Maria Oquendo, MD, Conte Center for the Neuroscience of Mental Disorders (CCNMD), New York State Psychiatric Institute, 1051 Riverside Drive, New York, NY, 10032. (Oquendo M. A., Halberstam B. & Mann J. J., Risk factors for suicidal behavior: utility and limitations of research instruments. In M.B. First [Ed.] Standardized Evaluation in Clinical Practice, pp. 103-130, 2003.)

For reprints of the C-SSRS contact Kelly Posner, Ph.D., New York State Psychiatric Institute, 1051 Riverside Drive, New York, New York, 10032; inquiries and training requirements contact posnerk@nyspi.columbia.edu

© 2008 The Research Foundation for Mental Hygiene, Inc

© 2008 Research Foundation for Mental Hygiene, Inc.

C-SSRS—Baseline/Screening (Version 1/14/09)

| SUICIDAL IDEATION | | | | | |
|---|---|---|---|---|---|
| Ask questions 1 and 2. If both are negative, proceed to "Suicidal Behavior" section. If the answer to question 2 is "yes", ask questions 3, 4 and 5. If the answer to question 1 and/or 2 is "yes", complete "Intensity of Ideation" section below. | | | Lifetime: Time<br>He/She Felt<br>Most Suicidal | | Past 6<br>Months |
| 1. Wish to be Dead Subject endorses thoughts about a wish to be dead or not alive anymore, or wish to fall asleep and not wake up. Have you wished you were dead or wished you could go to sleep and not wake up? | | Yes | No | Yes | No |
| If yes, describe: | | | | | |
| 2. Non-Specific Active Suicidal Thoughts General non-specific thoughts of wanting to end one's life/commit suicide (e.g., "Tve thought about killing myself") without thoughts of ways to kill oneself'associated methods, intent, or plan during the assessment period. Have you actually had any thoughts of killing yourself? If yes, describe: | | Yes | No | Yes | No |
| 3. Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act Subject endorses thoughts of suicide and has thought of at least one method during the assessment period. This is different than a specific plan with time, place or method details worked out (e.g., thought of method to kill self but not a specific plan). Includes person who would say, "I thought about taking an overdose but I never made a specific plan as to when, where or how I would actually do it and I would never go through with it." Have you been thinking about how you might do this? If yes, describe: | | Yes | No | Yes | No |
| 4. Active Suicidal Ideation with Some Intent to Act, without Specific Plan Active suicidal thoughts of killing oneself and subject reports having some intent to act on such thoughts, as opposed to "I have the thoughts but I definitely will not do anything about them." Have you had these thoughts and had some intention of acting on them? If yes, describe: | | Yes | No | Yes | No |
| 5. Active Suicidal Ideation with Specific Plan and Intent<br>Thoughts of killing oneself with details of plan fully or partially worked out and subject has some intent to carry it out.<br>Have you started to work out or worked out the details of how to kill yourself? Do you intend to carry out this plan? | | Yes | No | Yes | No |
| If yes, describe: | | | | | |
| INTENSITY OF IDEATION | | | | | |
| The following features should be rated with respect to the most severe type of ideation (i.e., 1-5 from above, with 1 being the least severe and 5 being the most severe). Ask about time he/she was feeling the most suicidal. | | | | | |
| Lifetime - Most Severe Ideation: Type # (1-5) | Description of Ideation | Most Severe Most<br>Severe | | | |
| Past 6 Months - Most Severe Ideation: Type # (1-5) | Description of Ideation | | | | |
| Frequency | Description of Insulan | | | | |
| How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in week (4) Daily or almost daily (5) Many times each day | | | _ | | _ |
| Duration | | | | | |
| When you have the thoughts how long do they last? (1) Fleeting - few seconds or minutes (2) Less than 1 hour/some of the time (3) 1-4 hours/a lot of time (5) More than 8 h | st of day<br>ours/persistent or continuous | _ | | _ | |
| Controllability Could/can you stop thinking about killing yourself or wanting to die if you want to? (1) Easily able to control thoughts (2) Can control thoughts with little difficulty (3) Unable to control thoughts | | | | _ | |
| (3) Can control thoughts with some difficulty (0) Does not atter | npt to control thoughts | | | | |
| Are there things - anyone or anything (e.g., family, religion, pain of death) - that stopped you from wanting to die or acting on thoughts of committing suicide? | | | | | |
| | st likely did not stop you<br>initely did not stop you<br>y | _ | | | _ |
| Reasons for Ideation What sort of reasons did you have for thinking about wanting to die or killing yourself? Was it to end the pain or stop the way you were feeling (in other words you couldn't go on living with this pain or how you were feeling) or was it to get attention, revenge or a reaction from others? Or both? (1) Completely to get attention, revenge or a reaction from others (2) Mostly to get attention, revenge or a reaction from others (3) Equally to get attention, revenge or a reaction from others and to end/stop the pain (5) Completely to end or stop the pain (you couldn't go on living with the pain or how you were feeling) (6) Completely to end or stop the pain (you couldn't go on living with the pain or how you were feeling) (9) Does not apply | | _ | | _ | |

© 2008 Research Foundation for Mental Hygiene, Inc.

C-SSRS—Baseline/Screening (Version 1/14/09)
| SUICIDAL BEHAVIOR (Check all that apply, so long as these are separate events; must ask about all types) | Life | time | Past<br>Yea | _ | |
|---|---|---|---|---|---|
| Actual Attempt: A potentially self-injurious act committed with at least some wish to die, as a result of act. Behavior was in part thought of as noneself. Intent does not have to be 100%. If there is any intent/desire to die associated with the act, then it can be considered an attempt. There does not have to be any injury or harm, just the potential for injury or harm. If person pulls trigger who mouth but gum is broken so no injury results, this is considered an attempt. Inferring Intent: Even if an individual denies intent/wish to die, it may be inferred clinically from the behavior or circumstances. | Yes | No | Yes | No | |
| a highly lethal act that is clearly not an accident so no other intent but suicide can be inferred (e.g., gunshot to head, jumping fiv<br>a highly lethal act that is clearly not an accident so no other intent but suicide can be inferred (e.g., gunshot to head, jumping fiv<br>a highly floor/story). Also, if someone demies intent to die, but they thought that what they did could be lethal, intent may be infer<br>Have you made a suicide attempt?<br>Have you done anything to harm yourself? | m window of | | | | |
| Have you done anything dangerous where you could have died? What did you do? | | | l#of<br>mpts | Total<br>Atter | |
| Did youas a way to end your life? Did you want to die (even a little) when you? Were you trying to end your life when you? Or did you think it was possible you could have died from? Or did you do it purely for other reasons / without ANY intention of killing yourself (like to relieve stress | feel hetter. | _ | _ | _ | _ |
| get sympathy, or get something else to happen)? (Self-Injurious Behavior without suicidal intent) If yes, describe: | , yeer sener, | Yes | No | Yes | No |
| Has subject engaged in Non-Suicidal Self-Injurious Behavior? | | | | | |
| Interrupted Attempt: When the person is interrupted (by an outside circumstance) from starting the potentially self-injurious act (if not for that, actual would have occurred). | l attempt | Yes | No | Yes | No |
| Overdose: Person has pills in hand but is stopped from ingesting. Once they ingest any pills, this becomes an attempt rather that attempt. Shooting: Person has gun pointed toward self, gun is taken away by someone else, or is somehow prevented from pulli. Once they pull the trigger, even if the gun fails to fire, it is an attempt. Jumping: Person is poised to jump, is grabbed and taken ledge. Hanging: Person has noose around neck but has not yet started to hang - is stopped from doing so. | | l#of | | | |
| Has there been a time when you started to do something to end your life but someone or something stopped you before you actually did anything? If yes, describe: | | | | Total | |
| Aborted Attempt: | | Yes | No | Yes | No |
| When person begins to take steps toward making a suicide attempt, but stops themselves before they actually have engaged in a destructive behavior. Examples are similar to interrupted attempts, except that the individual stops him/herself, instead of being something else. | stopped by | | | | |
| Has there been a time when you started to do something to try to end your life but you stopped yourself b actually did anything? If yes, describe: | efore you | | l#of<br>ated | Total<br>abor | |
| Preparatory Acts or Behavior: | | | | | |
| Acts or preparation towards imminently making a suicide attempt. This can include anything beyond a verbalization or thought, assembling a specific method (e.g., buying pills, purchasing a gun) or preparing for one's death by suicide (e.g., giving things a suicide note). | | Yes | No | Yes | No |
| Have you taken any steps towards making a suicide attempt or preparing to kill yourself (such as collecting a gun, giving valuables away or writing a suicide note)? If yes, describe: | ng pills, | | | | |
| Suicidal Behavior: Suicidal behavior was present during the assessment period? | | Yes | No | Yes | No |
| Answer for Actual Attempts Only | Most Recent<br>Attempt<br>Date: | Most Le<br>Attempt<br>Date: | ethal | Initial/Fi<br>Attempt<br>Date: | irst |
| Actual Lethality/Medical Damage: 0. No physical damage or very minor physical damage (e.g., surface scratches). | Enter Code | Enter | Code | Enter ( | Code |
| Minor physical damage (e.g., lethargic speech; first-degree burns; mild bleeding; sprains). Moderate physical damage; medical attention needed (e.g., conscious but sleepy, somewhat responsive; second-degree burns; bleeding of major vessel). | | | | | |
| <ol> <li>Moderately severe physical damage; medical hospitalization and likely intensive care required (e.g., comatose with reflexes intact; third-degree burns less than 20% of body; extensive blood loss but can recover; major fractures).</li> <li>Severe physical damage; medical hospitalization with intensive care required (e.g., comatose without reflexes; third- degree burns over 20% of body; extensive blood loss with unstable vital signs; major damage to a vital area).</li> <li>Death</li> </ol> | | _ | - | | _ |
| Detential Lethality: Only Answer if Actual Lethality=0 Likely lethality of actual attempt if no medical damage (the following examples, while having no actual medical damage, had potential for very serious lethality: put gun in mouth and pulled the trigger but gun fails to fire so no medical damage; laying on train tracks with oncoming train but pulled away before run over). | Enter Code | Enter | Code | Enter ( | Code |
| 0 = Behavior not likely to result in injury 1 = Behavior likely to result in injury but not likely to cause death 2 = Behavior likely to result in death despite available medical care | | _ | - | _ | _ |

© 2008 Research Foundation for Mental Hygiene, Inc.

C-SSRS—Baseline/Screening (Version 1/14/09)

#### 15.2.2. Since Last Visit Version

# COLUMBIA-SUICIDE SEVERITY RATING SCALE (C. SCRC)

(C-SSRS)

Since Last Visit

Version 1/14/09

Posner, K.; Brent, D.; Lucas, C.; Gould, M.; Stanley, B.; Brown, G.; Fisher, P.; Zelazny, J.; Burke, A.; Qquendo, M.; Mann, J.

#### Disclaimer:

This scale is intended to be used by individuals who have received training in its administration. The questions contained in the Columbia-Suicide Severity Rating Scale are suggested probes. Ultimately, the determination of the presence of suicidal ideation or behavior depends on the judgment of the individual administering the scale.

Definitions of behavioral suicidal events in this scale are based on those used in <u>The Columbia Suicide History Form</u>, developed by John Mann, MD and Maria <u>Oquendo</u>, MD, Conte Center for the Neuroscience of Mental Disorders (CCNMD), New York State Psychiatric Institute, 1051 Riverside Drive, New York, NY, 10032. (<u>Oquendo M. A., Halberstam</u> B. & Mann J. J., Risk factors for suicidal behavior: utility and limitations of research instruments. In M.B. First [Ed.] Standardized Evaluation in Clinical Practice, pp. 103-130, 2003.)

For reprints of the C-SSRS contact Kelly Posner, Ph.D., New York State Psychiatric Institute, 1051 Riverside Drive, New York, New York, 10032; inquiries and training requirements contact posnerk@nyspi.columbia.edu

© 2008 The Research Foundation for Mental Hygiene, Inc.

C-SSRS Since Last Visit - United States/English - Mapj. C-88R8-8InceLastVisit\_AU5.1\_eng-U8orl.doc

| SUICIDAL IDEATION | | | |
|---|---|---|---|
| Ask questions 1 and 2. If both are negative, proceed to "Suic<br>ask questions 3, 4 and 5. If the answer to question 1 and/or 1 | | | Last<br>sit |
| Wish to be Dead Subject endorses thoughts about a wish to be dead or not alive anymore, or Have you wished you were dead or wished you could go to sleep and not to | | Yes | No |
| If yes, describe: | | | |
| 2. Non-Specific Active Suicidal Thoughts General non-specific thoughts of wanting to end one's life/commit suicide oneself/associated methods, intent, or plan during the assessment period Have you actually had any thoughts of killing your self? If yes, describe: | (e.g., "I've thought about killing myself") without thoughts of ways to kill | Yes | No |
| | d during the assessment period. This is different than a specific plan with time,<br>not a specific plan). Includes person who would say, "I thought about taking an | Yes | No |
| 4. Active Suicidal Idea tion with Some Intent to Act, withou Active suicidal thoughts of killing oneself and subject reports having some will not do anything about them". Have you had these thoughts and had some intention of acting on them? If yes, describe: | intent to act on such thoughts, as opposed to "I have the thoughts but I definitely | Yes | No |
| 5. Active Suicidal Ideation with Specific Plan and Intent Thoughts of killing oneself with details of plan fully or partially worked ou Have you started to work out or worked out the details of how to kill your If yes, describe: | | Yes | No |
| INTENSITY OF IDEATION | | | |
| and 5 being the most severe). Most Severe Ideation: | ere type of ideation (i.e., 1-5 from above, with 1 being the least severe | | ost<br>ese |
| Туре # (1-5) | Description of Ideation | | |
| Frequency How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in weel | k (4) Daily or almost daily (5) Many times each day | | |
| Duration When you have the thoughts how long do they last? | | | |
| (1) Fleeting - few seconds or minutes<br>(2) Less than 1 hour/some of the time<br>(3) 1-4 hours/a lot of time | (4) 4-8 hours/most of day<br>(5) More than 8 hours/persistent or continuous | | _ |
| Controllability Could/can you stop thinking about killing yourself or wanting (1) Easily able to control thoughts (2) Can control thoughts with little difficulty (3) Can control thoughts with some difficulty | q to dis if you want to? (4) Can control thoughts with a lot of difficulty (5) Unable to control thoughts (0) Does not attempt to control thoughts | | _ |
| Deterrents | ain of death) - that stopped you from wanting to die or acting on | | |
| thoughts of committing suicide? | ainoj aeainj-inai sioppeayou jrom waraing to ale or acting on | | |
| (1) Deterrents definitely stopped you from attempting suicide (2) Deterrents probably stopped you (3) Uncertain that deterrents stopped you (0) Does not apply | | | |
| Reasons for Ideation | ** | | |
| What sort of reasons did you have for thinking about wanting you were feeling (in other words you couldn't go on living wit | to die or killing yourself? Was it to end the pain or stop the way<br>th this pain or how youwere feeling) or was it to get attention. | | |
| (1) Completely to get attention, revenge or a reaction from others (2) Mostly to get attention, revenge or a reaction from others (3) Mostly to get attention, revenge or a reaction from others (3) Equally to get attention, revenge or a reaction from others and to end/stop the pain | (4) Mostly to end or stop the pain (you couldn't go on living with the pain or how you were feeling) (5) Completely to end or stop the pain (you couldn't go on living with the pain or how you were feeling) (0) Does not apply | | |

| SUICIDAL BEHAVIOR | Since |
|---|---|
| (Check all that apply, so long as these are separate events; must ask about all types) | Last Visit |
| Actual Attempt: A potentially self-injurious act committed with at least some wish to die, as a result of act. Behavior was in part thought of as method to kill oneself. Intent does not have to be 100%. If there is any intent desire to die associated with the act, then it can be considered an actual suicide attempt. There does not have to be any injury or harm, just the potential for injury or harm. If person pulls trigger while gun is in mouth but gun is broken so no injury results, this is considered an attempt. | Yes No |
| Inferring Intent: Even if an individual denies intent/wish to die, it may be inferred clinically from the behavior or circumstances. For example, a highly lethal act that is clearly not an accident so no other intent but suicide can be inferred (e.g., gunshot to head jumping from window of a high floor/story). Also, if someonedenies intent to die, but they thought that what they did could be lethal, intent may be inferred. Have you made a suicide attempt? | |
| Have you done anything to harm yourself? Have you done anything dangerous where you could have died? What did you do? | Total # of<br>Attempts |
| Did you as a way to end your life? | Attempts |
| Did you want to die (even a little) when you? Were you trying to end your life when you? Or Did you think it was possible you could have died from? | |
| Or did you do it purely for other reasons / without ANY intention of killing yourself (like to relieve stress, feel better, get sympathy, or get something else to happen)? (Self-Injurious Behavior without suicidal intent) If yes, describe: | |
| Has subject engaged in Non-Suicidal Self-Injurious Behavior? | Yes No |
| Interrupted Attempt: | |
| When the person is interrupted (by an outside circumstance) from starting the potentially self-injurious act (if not for that, actual attempt would have occurred). Overdose: Person has pills in hand but is stopped from ingesting. Once they ingest any pills, this becomes an attempt rather than an interrupted attempt. Shooting: Person has gun pointed toward self, gun is taken away by someone else, or is somehow prevented from pulling trigger. Once they pull the trigger, even if the gun fails to fre, it is an attempt Jumping. Person is poised to jump, is grabbed and taken down from ledge. Hanging: Person has noose around neck but has not yet started to hang - is stopped from doing so. | Yes No |
| Has there been a time when you started to do something to end your life but someone or something stopped you before you actually did anything? If yes, describe: | Total # of<br>interrupted |
| n yes, describe. | |
| Aborted Attempt: When person begins to take steps toward making a suicide attempt, but stops themselves before they actually have engaged in any self-destructive behavior. Examples are similar to interrupted attempts, except that the individual stops him/herself, instead of being stopped by something else. Has there been a time when you started to do something to try to end your life but you stopped yourself before you actually did anything? If yes, describe: | Yes No Total # of aborted |
| Preparatory Acts or Behavior: Acts or preparation towards imminently making a suicide attempt. This can include anything beyond a verbalization or thought, such as assembling a specific method (e.g., buying pills, purchasing a gun) or preparing for one's death by suicide (e.g., giving things away, writing a suicide note). Have you taken any steps towards making a suicide attempt or preparing to kill yourself (such as collecting pills, getting a gun, giving valuables away or writing a suicide note)? If yes, describe: | Yes No |
| Suicidal Behavior:<br>Suicidal behaviorwas present during the assessment period? | Yes No |
| Suicide: | Yes No |
| Answer for Actual Attempts Only | Most Lethal<br>Attempt<br>Date: |
| Actual Lethality/Medical Damage: 0. No physical damage or very minor physical damage (e.g., surface scratches). | Enter Code |
| <ol> <li>Ninor physical damage (e.g., lethargic speech, first-degree burns; mild bleeding, sprains).</li> <li>Moderate physical damage; medical attention needed (e.g., conscious but sleepy, somewhat responsive; second-degree burns; bleeding of major vessel).</li> <li>Moderately severe physical damage; medical hospitalization and likely intensive care required (e.g., comatose with reflexes intact, third-degree burns less than 20% of body; extensive blood loss but can recover; major fractures).</li> <li>Severe physical damage; medical hospitalization with intensive care required (e.g., comatose without reflexes; third-degree burns over 20% of body; extensive blood loss with unstable vital signs; major damage to a vital area).</li> <li>Death</li> </ol> | |
| PotentialLethality: Only Answer if ActualLethality=0 | Enter Code |
| Likely leshality of actual attempt if no medical damage (the following examples, while having no actual medical damage, had potential for very serious leshality: put gun in mouth and pulled the trigger but gun fails to fire so no medical damage; laying on train tracks with oncoming train but pulled away before run over). | |
| 0 = Behavior not likely to result in injury 1 = Behavior likely to result in injury but not likely to cause death 2 = Behavior likely to result in death despite available medical care | |

# 15.3. Headache Impact Test (HIT-6 v1.0)

| HIT-6 <sup>TM</sup> | | HEADACHE IMPACT TEST | | |
|---|---|---|---|---|
| | This questionnaire was designed to help you describe and communicate the way you feel and what you cannot do because of headaches. | | | |
| To complete, please ch | To complete, please check one box for each question. | | | |
| 1. When you have head | laches, how often i | is the pain severe? | | |
| Never | Rarely | ☐ Sometimes | ☐ Very Often | Always |
| | 2. How often do headaches limit your ability to do usual daily activities including household work, work, school, or social activities? | | | |
| Never | Rarely | ☐ Sometimes | Very Often | Always |
| 3. When you have a he | adache, how often | do you wish you cou | ld lie down? | |
| Never | Rarely | ☐ Sometimes | ☐ Very Often | Always |
| 4. In the past 4 weeks, headaches? | how often have yo | u felt too tired to do v | vork or daily activition | es because of your |
| Never | Rarely | ☐ Sometimes | Very Often | Always |
| 5. In the past 4 weeks, how often have you felt fed up or irritated because of your headaches? | | | | |
| Never | Rarely | ☐ Sometimes | ☐ Very Often | Always |
| 6. In the past 4 weeks, how often did headaches limit your ability to concentrate on work or daily activities? | | | | |
| ■ Never | Rarely | Sometimes | ☐ Very Often | ☐ Always |

Headache Impact Test\*\* (HIT-6\*\*) © 2001, 2015 QualityMetric Incorporated and the GlaxoSmithKline Group of Companies. All rights reserved HIT-6\*\* United States (English) Version

### 15.4. Short-Form Health Survey (SF-36 v2.0)

1) In general, would you say your health is:

Very good

Excellent

#### Sample Short-Form Health Survey (SF-36 v2.0)

This survey asks for your views about your health. This information will help you keep track of how you feel and how well you are able to do your usual activities.

Please answer every question. Some questions may look like others, but each one is different. Please take the time to read and answer each question carefully, and click on the circle that best describes your answer. *Thank you for completing this survey!* 

Good

Fair

Poor

| | , , | | | |
|---|---|---|---|---|
| • | • | • | • | • |
| 2) Compared to or | ne year ago, how w | ould you rate your | health in generalno | <u>w</u> ? |
| Much better now than one year ago | Somewhat better<br>now than one<br>year ago | About the same as one year ago | Somewhat worse<br>now than one<br>year ago | Much worse now<br>than one year<br>ago |
| • | • | • | • | • |
| | | | you might do dur<br>s? If so, how mu | ring a typical day. |
| - | | Yes,<br>limited<br>a lot | Yes,<br>limited<br>a little | No, not<br>limited<br>at all |
| | <u>ties</u> , such as runni<br>ojects, participating<br>ts | | • | • |
| | <u>ities,</u> such as movi<br>g a vacuum cleane<br>ying golf | | • | • |
| c. Lifting or carry | ing groceries | • | • | • |
| d. Climbing <u>sever</u> | al flights of stairs | • | • | • |
| e. Climbing <u>one</u> fl | ight of stairs | • | • | • |
| f. Bending, kneel | ing, or stooping | • | • | • |
| g. Walking <u>more t</u> | han a mile | • | • | • |
| h. Walking <u>severa</u> | l hundred yards | • | • | • |
| i. Walking <u>one hu</u> | <u>indred yards</u> | • | • | • |

j. Bathing or dressing yourself



4) During the <u>past 4 weeks</u>, how much of the time have you had any of the following problems with your work or other regular daily activities <u>as a result of your physical health?</u>

| | of the<br>time | of the<br>time | of the<br>time | of the<br>time | of the time |
|---|---|---|---|---|---|
| <ul> <li>a. Cut down on<br/>the <u>amount of time</u> you<br/>spent on work or other<br/>activities</li> </ul> | • | • | • | • | • |
| <ul> <li>b. <u>Accomplished less</u> than you would like</li> </ul> | • | • | • | • | • |
| <ul> <li>Were limited in<br/>the <u>kind</u> of work or<br/>other activities</li> </ul> | • | • | • | • | • |
| d. Had <u>difficulty</u> performing<br>the work or other<br>activities (for example,<br>it took extra effort) | • | • | • | • | • |

5) During the <u>past 4 weeks</u>, how much of the time have you had any of the following problems with your work or other regular daily activities <u>as a result of any emotional problems</u> (such as feeling depressed or anxious)?



6) During the <u>past 4 weeks</u>, to what extent has your physical health or emotional problems interfered with your normal social activities with family, friends, neighbors, or groups?

Not at all Slightly Moderately Quite a bit Extremely

| 7) How much bo | | _ | 70 | | |
|---|---|---|---|---|---|
| None<br>• | Very Mild<br>● | Mild<br>• | Moderate<br>• | Severe<br>• | Very Severe |
| During the <u>pa</u> work outside the | | | nterfere with yo | ur normal w | ork (including both |
| Not at all | A little bit | Moderat | ely Quit | e a bit | Extremely |
| • | • | • | • | | • |
| 9) These ques<br>you <u>during the</u><br>comes closest<br>the <u>past 4 wee</u> | past 4 weeks. to the way you | For each que | stion, please | give the or | e answer that |
| | All of<br>the time | Most of<br>the time | Some of<br>the time | A little the tim | |
| a. Did you feel<br>full of life? | | • | • | • | • |
| b. Have you<br>been very<br>nervous? | • | • | • | • | • |
| c. Have you<br>felt so down<br>in the<br>dumps that<br>nothing<br>could cheer<br>you up? | • | • | • | • | • |
| d. Have you<br>felt calm and<br>peaceful? | • | • | • | • | • |
| e. Did you<br>have a lot of<br>energy? | • | • | • | • | • |
| f. Have you<br>felt<br>downhearted<br>and<br>depressed? | • | • | • | • | • |
| g. Did you feel<br>worn out? | • | • | • | • | • |
| h. Have you<br>been happy? | • | • | • | • | • |
| . D.1 | | | | | |

i. Did you feel tired? 10) During the past 4 weeks, how much of the time has your physical health or emotional problems interfered with your social activities (like visiting friends, relatives, etc.)?

All of the time Most of the time Some of the time A little of the None of the time time

| 11) How TRUE or FALSE is each | of the follo | wing state | ements fo | r you? | |
|---|---|---|---|---|---|
| | Definitely true | Mostly<br>true | Don't<br>know | Mostly false | Definitely<br>false |
| a. I seem to get sick a little easier than other people | • | • | • | • | • |
| b. I am as healthy as anybody I know | • | • | • | • | • |
| c. I expect my health to get worse | • | • | • | • | • |
| d. My health is excellent | _ | _ | _ | _ | |

## 15.5. Health Related Quality of Life (EQ-5D-5L)



**Health Questionnaire** 

English version for the USA

USA (English) © 2009 EuroQol Group EQ-5D™ is a trade mark of the EuroQol Group

| Under each heading, please check the ONE box that best describ | es your health TODAY. |
|---|---|
| MOBILITY | |
| I have no problems walking | |
| I have slight problems walking | |
| I have moderate problems walking | |
| I have severe problems walking | |
| I am unable to walk | |
| SELF-CARE | |
| I have no problems washing or dressing myself | |
| I have slight problems washing or dressing myself | |
| I have moderate problems washing or dressing myself | |
| I have severe problems washing or dressing myself | |
| I am unable to wash or dress myself | |
| USUAL ACTIVITIES (e.g. work, study, housework, family or leisure activities) | |
| I have no problems doing my usual activities | |
| I have slight problems doing my usual activities | |
| I have moderate problems doing my usual activities | |
| I have severe problems doing my usual activities | |
| I am unable to do my usual activities | |
| PAIN / DISCOMFORT | |
| I have no pain or discomfort | |
| I have slight pain or discomfort | |
| I have moderate pain or discomfort | |
| I have severe pain or discomfort | |
| I have extreme pain or discomfort | |
| ANXIETY / DEPRESSION | |
| I am not anxious or depressed | |
| I am slightly anxious or depressed | |
| I am moderately anxious or depressed | |
| I am severely anxious or depressed | |
| I am extremely anxious or depressed | |

2

USA (English) © 2009 EuroQol Group EQ-5D™ is a trade mark of the EuroQol Group

- We would like to know how good or bad your health is TODAY.
- . This scale is numbered from 0 to 100.
- 100 means the <u>best</u> health you can imagine.
   0 means the <u>worst</u> health you can imagine.
- Mark an X on the scale to indicate how your health is TODAY.
- Now, please write the number you marked on the scale in the box below.

YOUR HEALTH TODAY =

3

USA (English) © 2009 EuroQol Group EQ-5D™ is a trade mark of the EuroQol Group

# 15.6. Patient Global Impression of Change (PGIC)

| ratient Global Impression of Change (FGIC) | | | | |
|---|---|---|---|---|
| This section to be con | mpleted by site s | taff | | |
| Protocol: ALD403-C | LIN-011 | Subject #: | Visit Date | e: |
| Visit (please check or | ne): | | | |
| □ Week 4 | □ Week 8 | □ Week 12 | □ Week 16 | □ Week 20 |
| □ Week 24 | ☐ Week 32 or | ET | | |
| | MPTOMS, EMO | s study, how would you<br>OTIONS and OVERALL | | |
| Very Much Impr | roved | | | |
| Much Improved | | | | |
| Minimally Impro | oved | | | |
| No Change | | | | |
| Minimally Worse | е | | | |
| Much Worse | | | | |
| Very Much Wor | se | | | |

Version Date: 16 Aug 2016

## 15.7. Most Bothersome Symptom (MBS)

Most Bothersome Symptom (MBS)

| This section to be completed by site staff at each visit, Screening through Week 32 | | | | |
|---|---|---|---|---|
| Protocol: ALD403-C | LIN-011 St | ubject #: | Visit Date: _ | |
| Visit (please check or | ne): | | | |
| □ Screen | □ Day 0 | □ Week 4 | □ Week 8 | □ Week 12 |
| □ Week 16 | □ Week 20 | □ Week 24 | ☐ Week 32 or ET | |
| Most Bothersome Sy | mptom (as noted 1 | by subject at screening vi | sit): | |
| This section to be con | npleted by subject | at each visit, Day 0 throu | igh Week 32 | |
| Since beginning this symptom? Choose O | | you describe the change ( | if any) in your most bot | thersome |
| Very Much Impr | oved | | | |
| Much Improved | | | | |
| Minimally Impro | oved | | | |
| No Change | | | | |
| Minimally Worse | | | | |
| Much Worse | | | | |
| Very Much Worse | | | | |

Version Date: 17 Aug 2016

#### 15.8. References

- 1. Lipton R, Bigal M, Diamond M, Freitag F, Reed M, Stewart W. Migraine prevalence, disease burden, and the need for preventive therapy. Neurology. 2007; 68:343-349.
- 2. Leonardi M, Steiner TJ, Scher AT, Lipton RB. The global burden of migraine: measuring disability in headache disorders with WHO's classification of functioning, disability and health (ICF). J Headache Pain. 2005; 6(6):429-440.
- 3. Stewart WF, Ricci JA, Chee E, et al. Lost productive work time costs from health conditions in the United States: results from the American Productivity Audit J Occup Environ Med 2003; 45(12): 1234-1246.
- 4. Headache Classification Committee of the International Headache Society. The International Classification of Headache Disorders, 3rd edition (beta version). Cephalalgia. 2013:33(9):629-808.
- 5. Katsarava, Buse D. Defining differences between episodic and chronic migraine. Curr Pain and Headache. 2012; 1:86-92.
- 6. Buse DC, Manack A, Serrano D, Turkel C, Lipton RB. Sociodemographic and comorbidity profiles of chronic migraine and episodic migraine sufferers. J Neurol Neurosurg Psychiatry. 2010; 81 (4):428-432.
- 7. Durham PL. CGRP-receptor antagonists—a fresh approach to migraine therapy? N Engl J Med. 2004; 350:1073-1075.
- 8. Cady RJ, Shade CL, Cady RK. Advances in drug development for acute migraine. Drugs. 2012:72(17):1-19.
- 9. Durham PL. Calcitonin gene-related peptide (CGRP) and migraine. Headache. 2006; 46(Suppl 1):S3-S8.
- 10. Hansen JM, Hauge AW, Olesen J, Ashina M. Calcitonin gene-related peptide triggers migraine-like attacks in patients with migraine with aura. Cephalalgia. 2010; 30(10):1179-1186.
- 11. Schmid CW, Konrad M, Schmid DM, et al. the Journal of Headache and Pain 2013; 14:4
- 12. World Health Organization. International Classification of Diseases (ICD). Retrieved 23 Nov 2010.
- 13. United States Food and Drug Administration, United States Department of Health and Human Services. Guidance for Industry: Suicidal Ideation and Behavior: Prospective Assessment of Occurrence in Clinical Trials, Draft Guidance. August 2012. Revision 1.
- 14. Hintze, J. (2008) PASS 2008. NCSS, LLC. Kaysville, Utah. www.ncss.com
- LaVange L, Durham T, Koch G. Randomization-based Nonparametric Methods for the Analysis of Multicenter Trials. Statistical Methods in Medical Research. 2005; 14:281-301.
- 16. Mallinckrodt, C., Lipkovich, I. (2016). Analyzing Longitudinal Clinical Trial Data: A Practical Guide. Chapman and Hall/CRC Press, New York.

- 17. Esternalik E, Tepper S. Preventive treatment in migraine and the new US guidelines. Neuropsychiatr Dis Treat. 2013; 9; 709-720.
- 18. Antonaci F, Dumitrache C, De Cillis I, Allena M. A review of current European treatment guidelines for migraine. J Headache Pain. 2010; 11: 13-19.
- 19. Pringsheim T, Davenport W, Mackie G, et al. Canadian Headache Society Guideline for Migraine Prophylaxis Section II. Can J Neurol Sci 2012; 39: Suppl. 2 S8-28.